Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) – Amiloride vs Triamterene

NCT05125237

July 11, 2022

### 1. Comparison Details

### a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>amiloride versus triamterene</u> for hypertension.

### b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

### 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

### 3. Data Source(s)

Medicare, 2008-2018

### 4. Study Design Diagrams





### 5. Cohort Identification

### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing amiloride to triamterene. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of amiloride or triamterene (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

### b. Key details regarding cohort creation

#### Index date:

Day of initiation of new amiloride or triamterene use

### Inclusion criteria for analyses 1, 3, 4:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of amiloride, triamterene any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least two claims with hypertension diagnosis recorded in 365 days prior to index date

### Inclusion criteria for analysis 2:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of amiloride, triamterene any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least two claims with hypertension diagnosis recorded in 365 days prior to index date
- 180-day continuous use of amiloride or triamterene starting on the index date

# c. Flowchart of the study cohort assembly

| 4,362,962<br>83,290<br>53,837<br>7,039 | 25,300,359<br>937,397<br>554,107<br>200,270 |
|---|---|
| 83,290<br>53,837 | 554,107<br>200,270 |
| 53,837 | 200,270 |
| | - |
| 7,039 | 102 221 |
| | 183,231 |
| | 183,228 |
| 435 | 173,793 |
| 033 | 164,760 |
| 328 | 156,432 |
| 69 | 155,963 |
| | 7,476 |
| | 148,487 |
| | 155,963 |
| ,3 | 35 |

## 6. Variables

## a. Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of amiloride

## Comparator:

Initiators of amiloride will be compared to initiators of triamterene

## b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes | Anxiety |
| Obesity | Bipolar disorder |
| Coronary artery disease | Schizophrenia |
| Depression | |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of hospitalizations |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of C-reactive protein tests ordered |
| Pneumococcal vaccination | Osteoporosis |
| Herpes zoster vaccination | Fractures |

| Bone mineral density test | Falls |
|-----------------------------------|----------------------------|
| Number of distinct generic agents | Use of supplemental oxygen |
| Number of emergency room visits | Combined comorbidity score |
| Number of outpatient visits | |

| Comedication use | |
|---|---|
| Lithium | Nitrates |
| Anti-epileptic mood stabilizers | Lipid lowering drugs |
| Anti-epileptics (other than mood stabilizers) | Non-insulin diabetes medications |
| Atypical antipsychotics | Insulin |
| Benzodiazepines | Antidepressants |
| Serotonin-norepinephrine reuptake Inhibitors | Typical antipsychotics |
| Selective serotonin reuptake inhibitors | Anticoagulants |
| Tricyclic antidepressants (TCAs) | Antiplatelet agents |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Chronic liver disease |
| Coronary artery disease | Asthma |
| Heart failure | Ischemic heart disease |
| Stroke or transient ischemic attack | Chronic obstructive pulmonary disease |
| Peripheral vascular disease | Malignancy |
| Hyperlipidemia | Drug or alcohol abuse or dependence |
| Renal dysfunction | Venous thromboembolism |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:

#### Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of amiloride and triamterene and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (amiloride and triamterene) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of amiloride and triamterene and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

# 7. Feasibility counts

| Analysis scheme | Total amiloride/triamterene initiators | N outcome | Dementia Rate per<br>1,000 person-years<br>(95% CI) | Follow-up time in days; Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 6,794 (4.6%)<br>140,336 (95.4%) | 2,048 | 15.85 (15.16, 16.53) | 114 [29, 385] |
| 2: 6 mo induction period, 'as started' | 2,984 (4.7%)<br>59,943 (95.3%) | 3,232 | 24.74 (23.89, 25.60) | 897 [427, 1,095] |
| 3: exclude 6 mo follow-up (symptoms to claims period) | 2,896 (4.8%)<br>57,475 (95.2%) | 1,278 | 15.28 (14.46, 16.13) | 303 [111, 697] |
| 4: Outcome Dx + Rx | 6,794 (4.6%)<br>140,336 (95.4%) | 596 | 4.58 (4.22, 4.95) | 115 [29, 387] |

### 8. Propensity score analysis

We will use a propensity-score (PS)¹-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.² Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,³ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁴

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>5</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>6</sup>

# a. PS distributions stratified by treatment group

# Pre-matching propensity score overlap:



## Post-matching propensity score overlap:



# b. Table for covariate balance

| | Unm | Unmatched | | | PS-Matched | |
|---|---|---|---|---|---|---|
| Variable | Amiloride<br>(N = 7,476) | Triamterene<br>(N = 148,487) | St. Diff | Amiloride<br>(N = 7,424) | Triamterene<br>(N = 7,424) | St. Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 74.00 (6.59) | 74.97 (7.12) | -0.14 | 74.02 (6.60) | 74.16 (6.67) | -0.02 |
| Gender, n (%) | | | | | | 0.00 |
| Male | 3,164 (42.3%) | 50,177 (33.8%) | 0.18 | 3,129 (42.1%) | 3,153 (42.5%) | -0.01 |
| Female | 4,312 (57.7%) | 98,310 (66.2%) | -0.18 | 4,295 (57.9%) | 4,271 (57.5%) | 0.01 |
| Race, n (%) | | | | | | |
| White | 6,177 (82.6%) | 114,883 (77.4%) | 0.13 | 6,132 (82.6%) | 6,126 (82.5%) | 0.00 |
| Black | 831 (11.1%) | 20,547 (13.8%) | -0.08 | 828 (11.2%) | 815 (11.0%) | 0.01 |
| Asian | 123 (1.6%) | 5,061 (3.4%) | -0.12 | 122 (1.6%) | 123 (1.7%) | -0.01 |
| Hispanic | 127 (1.7%) | 3,968 (2.7%) | -0.07 | 127 (1.7%) | 141 (1.9%) | -0.02 |
| Native American | 23 (0.3%) | 682 (0.5%) | -0.03 | 23 (0.3%) | 18 (0.2%) | 0.02 |
| Unknown | 68 (0.9%) | 736 (0.5%) | 0.05 | 67 (0.9%) | 65 (0.9%) | 0.00 |
| Region, n (%) | | | | | | |
| Northeast; n (%) | 1,510 (20.2%) | 19,882 (13.4%) | 0.18 | 1,491 (20.1%) | 1,510 (20.3%) | 0.00 |
| South; n (%) | 2,841 (38.0%) | 64,874 (43.7%) | -0.12 | 2,825 (38.1%) | 2,838 (38.2%) | 0.00 |
| Midwest; n (%) | 1,958 (26.2%) | 34,300 (23.1%) | 0.07 | 1,947 (26.2%) | 1,924 (25.9%) | 0.01 |
| West; n (%) | 1,167 (15.6%) | 29,431 (19.8%) | -0.11 | 1,161 (15.6%) | 1,152 (15.5%) | 0.00 |
| Calendar year of index date, n (%) | | | | | | |
| 2008 | 570 (7.6%) | 15,514 (10.4%) | -0.10 | 568 (7.7%) | 590 (7.9%) | -0.01 |
| 2009 | 491 (6.6%) | 13,691 (9.2%) | -0.10 | 490 (6.6%) | 498 (6.7%) | 0.00 |
| 2010 | 419 (5.6%) | 11,796 (7.9%) | -0.09 | 418 (5.6%) | 422 (5.7%) | 0.00 |
| 2011 | 412 (5.5%) | 8,794 (5.9%) | -0.02 | 408 (5.5%) | 437 (5.9%) | -0.02 |
| 2012 | 409 (5.5%) | 7,753 (5.2%) | 0.01 | 408 (5.5%) | 382 (5.1%) | 0.02 |

| 2013 | 1,084 (14.5%) | 23,687 (16.0%) | -0.04 | 1,079 (14.5%) | 1,027 (13.8%) | 0.02 |
|---|---|---|---|---|---|---|
| 2014 | 1,089 (14.6%) | 21,542 (14.5%) | 0.00 | 1,081 (14.6%) | 1,081 (14.6%) | 0.00 |
| 2015 | 905 (12.1%) | 18,135 (12.2%) | 0.00 | 898 (12.1%) | 898 (12.1%) | 0.00 |
| 2016 | 715 (9.6%) | 10,459 (7.0%) | 0.09 | 710 (9.6%) | 734 (9.9%) | -0.01 |
| 2017 | 667 (8.9%) | 8,571 (5.8%) | 0.12 | 655 (8.8%) | 654 (8.8%) | 0.00 |
| 2018 | 715 (9.6%) | 8,545 (5.8%) | 0.14 | 709 (9.6%) | 701 (9.4%) | 0.01 |
| Low income subsidy, n (%) | 1,531 (20.5%) | 38,476 (25.9%) | -0.13 | 1,525 (20.5%) | 1,504 (20.3%) | 0.00 |
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 5,932 (79.3%) | 112,021 (75.4%) | 0.09 | 5,890 (79.3%) | 5,865 (79.0%) | 0.01 |
| Obesity | 2,041 (27.3%) | 29,567 (19.9%) | 0.17 | 2,021 (27.2%) | 2,056 (27.7%) | -0.01 |
| Coronary artery disease | 3,182 (42.6%) | 51,568 (34.7%) | 0.16 | 3,146 (42.4%) | 3,140 (42.3%) | 0.00 |
| Depression | 1,205 (16.1%) | 20,980 (14.1%) | 0.06 | 1,192 (16.1%) | 1,187 (16.0%) | 0.00 |
| Anxiety | 1,141 (15.3%) | 20,229 (13.6%) | 0.05 | 1,125 (15.2%) | 1,127 (15.2%) | 0.00 |
| Bipolar disorder | 142 (1.9%) | 1,551 (1.0%) | 0.08 | 140 (1.9%) | 147 (2.0%) | -0.01 |
| Schizophrenia | 46 (0.6%) | 757 (0.5%) | 0.01 | 46 (0.6%) | 40 (0.5%) | 0.01 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 1,922 (25.7%) | 26,672 (18.0%) | 0.19 | 1,897 (25.6%) | 1,909 (25.7%) | 0.00 |
| Mammography, n (%) | 1,548 (20.7%) | 31,823 (21.4%) | -0.02 | 1,545 (20.8%) | 1,538 (20.7%) | 0.00 |
| Colonoscopy, n (%) | 1,013 (13.6%) | 16,240 (10.9%) | 0.08 | 1,007 (13.6%) | 997 (13.4%) | 0.01 |
| Fecal occult blood test, n (%) | 627 (8.4%) | 12,989 (8.7%) | -0.01 | 617 (8.3%) | 608 (8.2%) | 0.00 |
| Influenza vaccination, n (%) | 4,887 (65.4%) | 90,529 (61.0%) | 0.09 | 4,854 (65.4%) | 4,906 (66.1%) | -0.01 |
| Pneumococcal vaccination, n (%) | 2,180 (29.2%) | 30,591 (20.6%) | 0.20 | 2,162 (29.1%) | 2,171 (29.2%) | 0.00 |
| Number of distinct prescriptions, mean (SD) | 16.13 (7.16) | 13.50 (6.43) | 0.39 | 16.07 (7.13) | 16.02 (7.52) | 0.01 |
| Number of emergency room visits, mean (SD) | 1.08 (1.85) | 0.75 (1.45) | 0.20 | 1.07 (1.84) | 1.04 (1.75) | 0.02 |
| Number of outpatient visits, mean (SD) | 19.01 (19.03) | 15.39 (19.09) | 0.19 | 18.87 (18.76) | 19.02 (18.96) | -0.01 |
| Number of hospitalizations, mean (SD) | 0.79 (1.34) | 0.41 (0.86) | 0.34 | 0.77 (1.32) | 0.75 (1.26) | 0.02 |
| Number of physician office visits, mean (SD) | 6.16 (9.69) | 6.32 (12.54) | -0.01 | 6.16 (9.71) | 6.24 (9.15) | -0.01 |

| Number of C-reactive protein tests ordered, mean (SD) | 0.28 (0.92) | 0.23 (0.84) | 0.06 | 0.28 (0.93) | 0.28 (0.95) | 0.00 |
|---|---|---|---|---|---|---|
| Number of serum creatinine tests ordered, mean (SD) | 6.93 (6.71) | 3.70 (3.26) | 0.61 | 6.73 (6.16) | 6.73 (7.11) | 0.00 |
| Composite frailty score, mean (SD) | 0.21 (0.07) | 0.20 (0.06) | 0.15 | 0.21 (0.07) | 0.21 (0.06) | 0.00 |
| Osteoporosis, n (%) | 953 (12.7%) | 19,417 (13.1%) | -0.01 | 944 (12.7%) | 913 (12.3%) | 0.01 |
| Fractures, n (%) | 599 (8.0%) | 10,241 (6.9%) | 0.04 | 591 (8.0%) | 532 (7.2%) | 0.03 |
| Falls, n (%) | 393 (5.3%) | 6,804 (4.6%) | 0.03 | 389 (5.2%) | 367 (4.9%) | 0.01 |
| Use of supplemental oxygen, n (%) | 266 (3.6%) | 2,350 (1.6%) | 0.13 | 259 (3.5%) | 250 (3.4%) | 0.01 |
| Combined comorbidity score, mean (SD) | 5.75 (3.36) | 3.87 (2.53) | 0.63 | 5.70 (3.32) | 5.76 (3.43) | -0.02 |
| Comedication use, n (%) | | | | | | |
| Lithium | 64 (0.9%) | 182 (0.1%) | 0.11 | 62 (0.8%) | 69 (0.9%) | -0.01 |
| Anti-epileptic mood stabilizers | 108 (1.4%) | 2,009 (1.4%) | 0.00 | 107 (1.4%) | 125 (1.7%) | -0.02 |
| Anti-epileptics (other than mood stabilizers) | 1,419 (19.0%) | 25,511 (17.2%) | 0.05 | 1,405 (18.9%) | 1,415 (19.1%) | -0.01 |
| Atypical antipsychotics | 186 (2.5%) | 2,917 (2.0%) | 0.03 | 178 (2.4%) | 180 (2.4%) | 0.00 |
| Benzodiazepines | 1,189 (15.9%) | 19,877 (13.4%) | 0.07 | 1,177 (15.9%) | 1,143 (15.4%) | 0.01 |
| Serotonin-norepinephrine reuptake inhibitors | 436 (5.8%) | 7,163 (4.8%) | 0.04 | 433 (5.8%) | 406 (5.5%) | 0.01 |
| Selective serotonin reuptake inhibitors | 1,263 (16.9%) | 23,241 (15.7%) | 0.03 | 1,251 (16.9%) | 1,287 (17.3%) | -0.01 |
| Tricyclic antidepressants (TCAs) | 388 (5.2%) | 7,252 (4.9%) | 0.01 | 385 (5.2%) | 373 (5.0%) | 0.01 |
| Typical antipsychotics | 46 (0.6%) | 706 (0.5%) | 0.01 | 46 (0.6%) | 50 (0.7%) | -0.01 |
| Anticoagulants | 1,489 (19.9%) | 18,773 (12.6%) | 0.20 | 1,469 (19.8%) | 1,438 (19.4%) | 0.01 |
| Antiplatelet agents | 1,104 (14.8%) | 21,979 (14.8%) | 0.00 | 1,099 (14.8%) | 1,077 (14.5%) | 0.01 |
| Nitrates | 1,097 (14.7%) | 17,217 (11.6%) | 0.09 | 1,086 (14.6%) | 1,109 (14.9%) | -0.01 |
| Lipid lowering drugs | 5,135 (68.7%) | 101,226 (68.2%) | 0.01 | 5,098 (68.7%) | 5,163 (69.5%) | -0.02 |
| Non-insulin diabetes medications | 3,946 (52.8%) | 78,139 (52.6%) | 0.00 | 3,917 (52.8%) | 3,964 (53.4%) | -0.01 |
| Insulin | 1,759 (23.5%) | 21,849 (14.7%) | 0.23 | 1,736 (23.4%) | 1,801 (24.3%) | -0.02 |
| Antidepressants | 2,148 (28.7%) | 38,805 (26.1%) | 0.06 | 2,131 (28.7%) | 2,109 (28.4%) | 0.01 |

| Comorbid conditions, n (%) | | | | | | |
|---|---|---|---|---|---|---|
| Atrial fibrillation | 1,951 (26.1%) | 24,709 (16.6%) | 0.23 | 1,922 (25.9%) | 1,857 (25.0%) | 0.02 |
| Heart failure | 2,594 (34.7%) | 30,271 (20.4%) | 0.32 | 2,559 (34.5%) | 2,555 (34.4%) | 0.00 |
| Stroke or transient ischemic attack | 752 (10.1%) | 14,344 (9.7%) | 0.01 | 747 (10.1%) | 762 (10.3%) | -0.01 |
| Peripheral vascular disease | 1,446 (19.3%) | 24,806 (16.7%) | 0.07 | 1,433 (19.3%) | 1,422 (19.2%) | 0.00 |
| Hyperlipidemia | 6,382 (85.4%) | 126,178 (85.0%) | 0.01 | 6,336 (85.3%) | 6,369 (85.8%) | -0.01 |
| Renal dysfunction | 3,323 (44.4%) | 28,925 (19.5%) | 0.55 | 3,276 (44.1%) | 3,314 (44.6%) | -0.01 |
| Chronic liver disease | 1,243 (16.6%) | 10,218 (6.9%) | 0.30 | 1,217 (16.4%) | 1,206 (16.2%) | 0.01 |
| Asthma | 1,351 (18.1%) | 22,260 (15.0%) | 0.08 | 1,338 (18.0%) | 1,316 (17.7%) | 0.01 |
| Ischemic heart disease | 3,400 (45.5%) | 57,004 (38.4%) | 0.14 | 3,365 (45.3%) | 3,351 (45.1%) | 0.00 |
| Chronic obstructive pulmonary disease | 2,016 (27.0%) | 35,094 (23.6%) | 0.08 | 1,997 (26.9%) | 1,985 (26.7%) | 0.00 |
| Malignancy | 2,536 (33.9%) | 39,520 (26.6%) | 0.16 | 2,502 (33.7%) | 2,635 (35.5%) | -0.04 |
| Drug or alcohol abuse or dependence | 830 (11.1%) | 12,524 (8.4%) | 0.09 | 822 (11.1%) | 826 (11.1%) | 0.00 |
| Venous thromboembolism | 527 (7.0%) | 7,480 (5.0%) | 0.08 | 520 (7.0%) | 515 (6.9%) | 0.00 |

### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease. In addition to the Medicare dataset, we will pursue a similar analysis within Clinical Practice Research Datalink (CPRD), a UK population health dataset, to validate our results.

### 10. References

- 1. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 5. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. Comp Effect Res 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- **7.** Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.

| # | Implementation in routine care | |
|---|---|---|
| | EXPOSURE vs. COMPARISON | |
| | Amiloride vs Triamterene | |
| | INCLUSION CRITERIA | |
| 1 | Age | Aged > 65 years on the index date |
| | Hypertension diagnosis | Measured 365 days prior to drug initiation for at least two claims in any diagnosis position and inpatient or outpatient outpatient setting – |
| 2 | | ICD9 diagnosis – 401.1, 401.9, 402.10, 402.90, 404.10, 404.90, 405.11, 405.19, 405.91, 405.99<br>ICD10 diagnosis – 110-115.x, N26.2 |
| 3 | Sufficient enrollment | Medicare Part A, B, and D enrollment with no HMO coverage for 365 days prior to and on the cohort entry date |
| | | EXCLUSION CRITERIA |
| 1 | Prior history of dementia | Measured any time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – ICD9 diagnosis – 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 ICD10 diagnosis – F01.xx-F03.xx, G30.xx-G31.85, R41.xx NDC brand name – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or |
| | | "REMINYL" NDC generic name – "DONEPEZIL HCL", "GALANTAMINE HBR", "MEMANTINE HCL", "MEMANTINE HCL/DONEPEZIL HCL", "RIVASTIGMIN or "RIVASTIGMINE TARTRATE" |
| 2 | Prior use of study drugs | Measured any time prior to drug initiation – Amiloride Triamterene |

| Covariate list | |
|---|---|
| Category | Potential confounders |
| Category | ICD-9 |
| | Age |
| | Gender |
| Demographics | Race |
| | Region |
| | Calendar year of index date |
| | Low income subsidy |
| | 211 |
| | Diabetes |
| | Obesity |
| | Coronary artery disease |
| Dementia risk factors | Depression |
| | Anxiety |
| | Bipolar disorder |
| | Schizophrenia |
| | Const. |
| | Smoking |
| | Mammography |
| | Colonoscopy |
| Lifestyle factors and markers for healthy behavior | Fecal occult blood test |
| | Influenza vaccination |
| | Pneumococcal vaccination |
| | Herpes zoster vaccination |
| | BMD test |
| | No contract of distinct on a sign of a sector |
| | Number of distinct generic agents |
| | Number of emergency room visits |
| Healthcare utilization measures | Number of outpatient visits |
| ricalticale utilization measures | Number of hospitalizations |
| | Number of physician office visits Number of CRP tests ordered |
| | Number of ckr tests ordered Number of serum creatinine tests ordered |
| | Number of serum creatinine tests of dered |
| | Composite frailty score |
| | Osteoporosis |
| | Fractures |
| Frailty markers | Falls |
| | Use of supplemental oxygen |
| | A combined comorbidity score |
| | Accomplised complainty score |
| | Lithium |
| | Anti-epileptic mood stabilizers |
| | Anti-epileptics (other than mood stabilizers) |
| | Atypical antipsychotics |
| | Benzodiazepines |
| | Denzouluzepines |

| | SNRIs |
|---------------------|-------------------------------------|
| | SSRIs |
| Comedications | TCAs |
| Comedications | Typical antipsychotics |
| | Anticoagulants |
| | Antiplatelet agents |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Diabetes |
| | Hyperlipidemia |
| Comorbid conditions | Renal dysfunction |
| | Chronic liver disease |
| | Asthma |
| | Ischemic heart disease |
| | COPD |
| | Malignancy |
| | Drug or alcohol abuse or dependence |
| | VTE |

# Appendix A Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |
| 2018 |

### Low income subsidy

https://www.cms.gov/Medicare/Eligibility-and-Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pdf

### Diabetes


## Obesity


## Appendix A Dementia risk factors


Sibutramine
Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

Orlistat

Hypertension

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| I10 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| I10 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| I160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| I161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| I110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| I110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, malignant, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| l129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| I129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |

| 11311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
|---|---|---|---|
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | stage renal disease | or end stage renal disease |
| 11310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| 1130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| I1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| 1150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| 1158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| 1150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| 1151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| 1152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| 1158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| 1158 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |
| 1133 | 40333 | pecondary hypertension, unspecified | Totaler dispersified secondary hypertension |

onary artery disease


| 33519 |
|----------|
| 33520 |
| 33521 |
| 33522 |
| 33523 |
| 33524 |
| 33525 |
| 33526 |
| 33527 |
| 33528 |
| 33529 |
| 33530 |
| 33531 |
| 33532 |
| 33533 |
| 33534 |
| 33535 |
| 33536 |
| 33545 |
| 33572 |
| CPT |
| 92973 |
| 92982 |
| 92984 |
| 92995 |
| 92996 |
| 92920 |
| 92921 |
| 92924 |
| 92925 |
| 92937 |
| 92938 |
| 92941 |
| 92943 |
| 92944 |
| ICD10 Dx |
| 1200 |


| Dilation of Coronary Artery, Two Arteries with cronary artery stent(s) Dilation of Coronary Artery, Two Arteries, coronary artery stent(s) Dilation of Coronary Artery, Two Arteries, direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of direction of Dilation of Coronary Artery, Three Arteries, direction of Dilation of Coronary Artery, Three Arteries, direction of direction of direction of Dilation of Coronary Artery, Three Arteries direction of | luccution of | | 1 | |
|---|---|---|---|---|
| Three Drug-eluting Intraluminal Devices, coronary artery | Insertion of | Dilation of Caranagu Artagu Two Artarias with | | |
| Dilation of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries with a forum of Grown of Grown of Coronary Artery, Two Arteries with forum of Grown of More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal or Grown or Approach stent(s) Dilation of Coronary Artery, Three Arteries, and Grown or G | = = | · | | |
| Dilation of Coronary Artery, Two Arteries, dinsertion of Bifurcation, with Four or More Drug-eluting drug-eluting drug-eluting coronary artery stent(s) 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with Insertion of Grug-eluting Devices, Percutaneous Endoscopic coronary artery stent(s) 0271472 3607 Approach Significant of Coronary Artery, Two Arteries with Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) 0272046 3607 Device, Open Approach stent(s) 0272047 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272048 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery stent(s) 0272049 Significant of Coronary Artery, Three Arteries, drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272050 Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272051 Significant of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach Stent(s) 0272052 3607 Open Approach Significant of Coronary Artery, Three Arteries Sifurcation, with Twee Drug-eluting Coronary artery Stent(s) 0272066 3607 Significant of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) 0272067 Significant Sig | | , | 2607 | 0274467 |
| Bifurcation, with Four or More Drug-eluting coronary artery stent(s) 0271476 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) 0271472 3607 Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting moronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Fo | ` ' | | 3607 | 02/1462 |
| Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) | | · | | |
| Dilation of Coronary Artery, Three Arteries with Insertion of Grug-eluting Intraluminal Devices, Open Approach | 0 0 | , | | |
| Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary arte | | - | 2607 | 0274476 |
| Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting mornary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) | | | 3607 | 02/14/6 |
| Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | · | | |
| 027147Z 3607 Approach Stent(s) Insertion of drug-eluting coronary artery stent(s) O272046 3607 Device, Open Approach O272046 O272047 O272047 O272047 O272048 O | ŭ ŭ | | | |
| Dilation of Coronary Artery, Three Arteries, setults and setulting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, with Drug-eluting Intraluminal pevice, Open Approach Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) | | - | 2607 | 0274 477 |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Device, Open Approach Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries Bifurcation, with Three Drug-eluting Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Ar | ` ' | Approacn | 3607 | 02/14/2 |
| Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, or | | Dilation of Common Adam Thomas Adams | | |
| 0272046 3607 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting sention of Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting linsertion of linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting linsertion of drug-eluting linsertion of drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) | = = | · | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting gradient stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | ` ' | Device, Open Approach | 3607 | 0272046 |
| with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272052 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) | | | | |
| 0272042 3607 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, with Two Drug-eluting Intraluminal Devices, oronary artery 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 027206B 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, with Three Drug-eluting Coronary artery 027206C 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Coronary artery stent(s) Insertion of drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery Open | = = | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027207G 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027207G 3607 Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | ' ' | | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Insertion of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Stent(s) | | Approach | 3607 | 027204Z |
| Bifurcation, with Two Drug-eluting coronary artery stent(s) Section of Coronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries, and the section of drug-eluting loronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and the section of drug-eluting loronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and the section of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries and the section of drug-eluting loronary artery stent(s) Dilation of Coronary Artery, Three Arteries and the section of drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and the section of drug-eluting loronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and the section of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries and the section of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries and the section of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and the section of drug-eluting coronary artery stent section of drug-eluting coronary artery section of drug-eluting coronary artery stent section of drug-eluting coronary artery sect | | | | |
| 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) O27205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Three Drug-eluting coronary artery stent(s) O272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Dilation of Coronary Artery, Three Arteries drug-eluting 3607 Dilation of Coronary Artery, Three Arteries drug-eluting 3607 Dilation of Coronary Artery, Three Arteries drug-eluting 3607 Devices, Open Approach stent(s) 3607 Dilation of Coronary Artery, Three Arteries, drug-eluting 3607 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | | | |
| Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, stent(s) Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Oz72066 3607 Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Sifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Gronary Artery Stent(s) Insertion Of Gronary Artery Stent Stent(s) Insertion Of Gronary Artery Stent Stent(s) Insertion Of Gronary Artery Stent St | ` ' | Intraluminal Devices, Open Approach | 3607 | 0272056 |
| with Two Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, With Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Sifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | | | | |
| 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery with Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Insertion of drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery | | · | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z O27 | , coronary artery | with Two Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries With Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries With Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting O272076 3607 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries With Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries With Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries With Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | stent(s) | Open Approach | 3607 | 027205Z |
| Bifurcation, with Three Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Devices, Open Approach stent(s) | Insertion of | | | |
| 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 0272072 3607 Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 0272072 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting drug-eluting coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting coronary artery 027207Z Grid drug-eluting drug-eluting coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Four or More Drug-eluting coronary artery stent(s) O272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) O27207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Three Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery Bifurcation, with Four or More Drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, green of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | | Intraluminal Devices, Open Approach | 3607 | 0272066 |
| with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting | Insertion of | | | |
| 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting insertion of drug-eluting coronary artery coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z Graph Grap | es, coronary artery | with Three Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal 027207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Devices, Open Approach Insertion of drug-eluting drug-eluting drug-eluting coronary artery Coronary artery | stent(s) | Open Approach | 3607 | 027206Z |
| Bifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Insertion of drug-eluting coronary artery | Insertion of | | | |
| 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Four or More Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | stent(s) | Intraluminal Devices, Open Approach | 3607 | 0272076 |
| with Four or More Drug-eluting Intraluminal coronary artery 3607 Devices, Open Approach stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | 0 0 | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | l coronary artery | with Four or More Drug-eluting Intraluminal | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | Devices, Open Approach | 3607 | 027207Z |
| Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| | drug-eluting | | | |
| 0272346 3607 Device, Percutaneous Approach | coronary artery | Bifurcation, with Drug-eluting Intraluminal | | |
| Jeney | stent(s) | Device, Percutaneous Approach | 3607 | 0272346 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Drug-eluting Intraluminal Device, coronary artery | coronary artery | with Drug-eluting Intraluminal Device, | | |
| 027234Z 3607 Percutaneous Approach stent(s) | stent(s) | Percutaneous Approach | 3607 | 027234Z |
| Dilation of Coronary Artery, Three Arteries, Insertion of | Insertion of | Dilation of Coronary Artery, Three Arteries, | | |
| Bifurcation, with Two Drug-eluting drug-eluting | drug-eluting | Bifurcation, with Two Drug-eluting | | |
| Intraluminal Devices, Percutaneous coronary artery | coronary artery | Intraluminal Devices, Percutaneous | | |
| 0272356 3607 Approach stent(s) | stent(s) | Approach | 3607 | 0272356 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Two Drug-eluting Intraluminal Devices, coronary artery | | | | |
| 027235Z 3607 Percutaneous Approach stent(s) | | | 3607 | 027235Z |


## Depression


Anxiety


Bipolar disorder


Schizophrenia

# Appendix A Dementia risk factors


#### **Smoking**


CPT codes
99406
99407
G0436
G0437
G9016
S9453
S4995
G9276
G9458
1034F
4001F
4004F

OR dispensing of: At least one nicotine or varenicline prescription

#### Mammography


Colonoscopy


**CPT**45378
45379

# Appendix A Lifestyle factors and markers for healthy behavior

| 45380 |
|-------|
| 45381 |
| 45382 |
| 45383 |
| 45384 |
| 45385 |
| 45386 |
| 45387 |
| 45388 |
| 45389 |
| 45390 |
| 45391 |
| 45392 |
| HCPCS |
| G0105 |
| G0121 |

#### Fecal occult blood test


#### Influenza vaccination


| <b>U.</b> . |
|-------------|
| 90655 |
| 90656 |
| 90657 |
| 90658 |
| 90659 |
| 90660 |
| 90724 |
| HCPCS |
| G0008 |

#### Pneumococcal vaccination


# Appendix A Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

#### Herpes zoster vaccination

| - 1 |
|-------|
| CPT |
| 90376 |
| 90750 |

#### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

### Appendix A Healthcare utilization measures

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | HCPCS | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

#### Number of CRP tests

| CPT | |
|-------|-------|
| 86140 | 86141 |

#### Number of serum creatinine tests


# Appendix A Frailty markers

#### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| ntestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality<br>Disorders, And Other Nonpsychotic<br>Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.921, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | 130-139 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36 (excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

## Appendix A Frailty markers

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | \$81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

## Appendix A Frailty markers

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

## Appendix A Frailty markers

Osteoporosis

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDesICD9 |
|---|---|---|---|
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| e of thumb [first] metacarpal |
|-------------------------------------------|
| a of thumb [first] matagarnal |
| e of thumb [first] metacarpal |
| . , . |
| e of other metacarpal bone(s) |
| e of other metacarpal bone(s) |
| ft of metacarpal bone(s) |
| ft of metacarpal bone(s) |
| k of metacarpal bone(s) |
| k of metacarpal bone(s) |
| tiple sites of metacarpus |
| acarpal bone(s), site unspecified |
| of thumb [first] metacarpal |
| or triumb (iiist) metacarpar |
| of thumb [first] metacarpal |
| or triams (mot) metacarpar |
| of other metacarpal bone(s) |
| , |
| of other metacarpal bone(s) |
| of metacarpal bone(s) |
| of metacarpal bone(s) |
| of metacarpal bone(s) |
| of metacarpal bone(s) |
| iple sites of metacarpus |
| lanx or phalanges of hand, unspecified |
| ianx or pharanges of hand, unspecified |
| lanx or phalanges of hand, unspecified |
| ianix or priaranges or naria, anspectivea |
| dle or proximal phalanx or phalanges of |
| and an increase process of process of |
| dle or proximal phalanx or phalanges of |
| dle or proximal phalanx or phalanges of |
| dle or proximal phalanx or phalanges of |
| dle or proximal phalanx or phalanges of |
| al phalanx or phalanges of hand |
| al phalanx or phalanges of hand |
| al phalanx or phalanges of hand |
| al phalanx or phalanges of hand |
| ff ff k k t |


| 8250 | Salter-Harris Type III physeal fracture of unspecified | Fracture of calcaneus, closed |
|---|---|---|
| 8250 | Salter-Harris Type IV physeal fracture of unspecified calcaneus, initial encounter for closed fracture | Fracture of calcaneus, closed |
| 8250 | Other physeal fracture of unspecified calcaneus, initial | Fracture of calcaneus, closed |
| 8251 | Unspecified fracture of unspecified calcaneus, initial | Fracture of calcaneus, open |
| | encounter for open fracture | |
| 8251 | Unspecified physeal fracture of unspecified calcaneus, initial encounter for open fracture | Fracture of calcaneus, open |
| 8251 | Salter-Harris Type I physeal fracture of unspecified calcaneus, | Fracture of calcaneus, open |
| 8251 | Salter-Harris Type II physeal fracture of unspecified | Fracture of calcaneus, open |
| 8251 | | Fracture of calcaneus, open |
| | calcaneus, initial encounter for open fracture | |
| 8251 | Salter-Harris Type IV physeal fracture of unspecified calcaneus, initial encounter for open fracture | Fracture of calcaneus, open |
| 8251 | Other physeal fracture of unspecified calcaneus, initial | Fracture of calcaneus, open |
| 82520 | Other fracture of unspecified foot, initial encounter for closed | Closed fracture of unspecified bone(s) of foot [except toes] |
| 82520 | Unspecified fracture of unspecified foot, initial encounter for | Closed fracture of unspecified bone(s) of foot [except toes] |
| 82521 | Unspecified fracture of unspecified talus, initial encounter for | Closed fracture of astragalus |
| 02522 | closed fracture | Classed from the continuous for a contin |
| 82522 | initial encounter for closed fracture | Closed fracture of navicular [scaphoid], foot |
| 82522 | Nondisplaced fracture of navicular [scaphoid] of unspecified foot, initial encounter for closed fracture | Closed fracture of navicular [scaphoid], foot |
| 82523 | Displaced fracture of cuboid bone of unspecified foot, initial | Closed fracture of cuboid |
| 82523 | Nondisplaced fracture of cuboid bone of unspecified foot, | Closed fracture of cuboid |
| 82524 | Displaced fracture of lateral cuneiform of unspecified foot, | Closed fracture of cuneiform, foot |
| 82524 | | Closed fracture of cuneiform, foot |
| 82524 | initial encounter for closed fracture | Closed fracture of cuneiform, foot |
| 82324 | foot, initial encounter for closed fracture | closed if acture of currenorm, foot |
| 82524 | · · | Closed fracture of cuneiform, foot |
| 82524 | Displaced fracture of medial cuneiform of unspecified foot, | Closed fracture of cuneiform, foot |
| 82524 | Nondisplaced fracture of medial cuneiform of unspecified foot, | Closed fracture of cuneiform, foot |
| 82525 | Fracture of unspecified metatarsal bone(s), unspecified foot, | Closed fracture of metatarsal bone(s) |
| 82525 | initial encounter for closed fracture Unspecified physeal fracture of unspecified metatarsal, initial | Closed fracture of metatarsal bone(s) |
| | encounter for closed fracture | ., |
| | Salter-Harris Type I physeal fracture of unspecified metatarsal, initial encounter for closed fracture | Closed fracture of metatarsal bone(s) |
| 82525 | Salter-Harris Type II physeal fracture of unspecified metatarsal, initial encounter for closed fracture | Closed fracture of metatarsal bone(s) |
| 82525 | Salter-Harris Type III physeal fracture of unspecified | Closed fracture of metatarsal bone(s) |
| 82525 | Salter-Harris Type IV physeal fracture of unspecified | Closed fracture of metatarsal bone(s) |
| 82525 | | Closed fracture of metatarsal bone(s) |
| | encounter for closed fracture | |
| | 8250<br>8250<br>8251<br>8252<br>82520<br>82520<br>82520<br>82522<br>82522<br>82523<br>82524<br>82524<br>82524<br>82524<br>82524<br>82524<br>82525<br>82525<br>82525<br>82525 | calcaneus, initial encounter for closed fracture 8250 Salter-Harris Type IV physeal fracture of unspecified calcaneus, initial encounter for closed fracture 8250 Other physeal fracture of unspecified calcaneus, initial encounter for closed fracture 8251 Unspecified fracture of unspecified calcaneus, initial encounter for open fracture 8251 Unspecified physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Salter-Harris Type II physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Salter-Harris Type II physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Salter-Harris Type III physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Salter-Harris Type IV physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Salter-Harris Type IV physeal fracture of unspecified calcaneus, initial encounter for open fracture 8251 Other physeal fracture of unspecified calcaneus, initial encounter for open fracture 8252 Other fracture of unspecified foot, initial encounter for closed fracture 8252 Unspecified fracture of unspecified foot, initial encounter for closed fracture 8252 Unspecified fracture of unspecified foot, initial encounter for closed fracture 8252 Displaced fracture of navicular [scaphoid] of unspecified foot, initial encounter for closed fracture 8252 Nondisplaced fracture of navicular [scaphoid] of unspecified foot, initial encounter for closed fracture 8252 Nondisplaced fracture of cuboid bone of unspecified foot, initial encounter for closed fracture 8252 Nondisplaced fracture of intermediate cuneiform of unspecified foot, initial encounter for closed fracture 82524 Displaced fracture of intermediate cuneiform of unspecified foot, initial encounter for closed fracture 82524 Nondisplaced fracture of intermediate cuneiform of unspecified metatures of intermediate cuneiform of unspecified foot, initial encounter for closed fracture 82524 Nondisplaced |


| | _ | |
|---|---|---|
| 80607 | Unspecified nondisplaced fracture of seventh cervical | Closed fracture of C5-C7 level with anterior cord syndrome |
| 80607 | Anterior cord syndrome at C5 level of cervical spinal cord, | Closed fracture of C5-C7 level with anterior cord syndrome |
| 80607 | Anterior cord syndrome at C6 level of cervical spinal cord, | Closed fracture of C5-C7 level with anterior cord syndrome |
| 80607 | Anterior cord syndrome at C7 level of cervical spinal cord, | Closed fracture of C5-C7 level with anterior cord syndrome |
| 80608 | Unspecified displaced fracture of fifth cervical vertebra, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Unspecified nondisplaced fracture of fifth cervical vertebra, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Unspecified displaced fracture of sixth cervical vertebra, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Unspecified nondisplaced fracture of sixth cervical vertebra, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Unspecified displaced fracture of seventh cervical vertebra, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Unspecified nondisplaced fracture of seventh cervical | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | vertebra, initial encounter for closed fracture Central cord syndrome at C5 level of cervical spinal cord, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | initial encounter Central cord syndrome at C6 level of cervical spinal cord, | Closed fracture of C5-C7 level with central cord syndrome |
| 80608 | Central cord syndrome at C7 level of cervical spinal cord, | Closed fracture of C5-C7 level with central cord syndrome |
| 80609 | Unspecified displaced fracture of fifth cervical vertebra, | Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | Unspecified nondisplaced fracture of fifth cervical vertebra, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | Unspecified displaced fracture of sixth cervical vertebra, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | initial encounter for closed fracture Unspecified nondisplaced fracture of sixth cervical vertebra, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | initial encounter for closed fracture Unspecified displaced fracture of seventh cervical vertebra, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | initial encounter for closed fracture Unspecified nondisplaced fracture of seventh cervical | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | vertebra, initial encounter for closed fracture Other incomplete lesion at C5 level of cervical spinal cord, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | initial encounter Other incomplete lesion at C6 level of cervical spinal cord, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80609 | initial encounter Other incomplete lesion at C7 level of cervical spinal cord, | injury Closed fracture of C5-C7 level with other specified spinal cord |
| 80610 | initial encounter Unspecified displaced fracture of first cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture Unspecified nondisplaced fracture of first cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture Unspecified displaced fracture of second cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture Unspecified nondisplaced fracture of second cervical | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | vertebra, initial encounter for open fracture Unspecified displaced fracture of third cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture Unspecified displaced fracture of fourth cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| 80610 | initial encounter for open fracture Unspecified nondisplaced fracture of fourth cervical vertebra, | injury Open fracture of C1-C4 level with unspecified spinal cord |
| | 80607 80607 80607 80608 80608 80608 80608 80608 80608 80608 80609 | vertebra, initial encounter for closed fracture 80607 Anterior cord syndrome at C5 level of cervical spinal cord, initial encounter 80607 Anterior cord syndrome at C6 level of cervical spinal cord, initial encounter 80607 Anterior cord syndrome at C7 level of cervical spinal cord, initial encounter 80608 Unspecified displaced fracture of fifth cervical vertebra, initial encounter for closed fracture 80608 Unspecified nondisplaced fracture of fifth cervical vertebra, initial encounter for closed fracture 80608 Unspecified displaced fracture of sixth cervical vertebra, initial encounter for closed fracture 80608 Unspecified onodisplaced fracture of sixth cervical vertebra, initial encounter for closed fracture 80608 Unspecified onodisplaced fracture of seventh cervical vertebra, initial encounter for closed fracture 80608 Unspecified onodisplaced fracture of seventh cervical vertebra, initial encounter for closed fracture 80608 Central cord syndrome at C5 level of cervical spinal cord, initial encounter 80608 Central cord syndrome at C5 level of cervical spinal cord, initial encounter 80609 Unspecified displaced fracture of fifth cervical vertebra, initial encounter 80609 Unspecified onodisplaced fracture of fifth cervical vertebra, initial encounter 80609 Unspecified onodisplaced fracture of fifth cervical vertebra, initial encounter for closed fracture 80609 Unspecified onodisplaced fracture of sixth cervical vertebra, initial encounter for closed fracture 80609 Unspecified onodisplaced fracture of sixth cervical vertebra, initial encounter for closed fracture 80609 Unspecified onodisplaced fracture of sixth cervical vertebra, initial encounter for closed fracture 80609 Unspecified nondisplaced fracture of seventh cervical vertebra, initial encounter for closed fracture 80609 Unspecified nondisplaced fracture of seventh cervical vertebra, initial encounter for open fracture 80600 Unspecified nondisplaced fracture of first cervical vertebra, initial encounter for open fracture 80610 Unspecif |


| | | T |
|---|---|---|
| 8083 | Fracture of superior rim of left pubis, initial encounter for open fracture | Open fracture of pubis |
| 8083 | Fracture of superior rim of unspecified pubis, initial encounter for open fracture | Open fracture of pubis |
| 8083 | Other specified fracture of right pubis, initial encounter for | Open fracture of pubis |
| 8083 | Other specified fracture of left pubis, initial encounter for | Open fracture of pubis |
| 8083 | Other specified fracture of unspecified pubis, initial encounter | Open fracture of pubis |
| 80841 | Unspecified fracture of right ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | Unspecified fracture of left ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | Displaced avulsion fracture of right ilium, initial encounter | Closed fracture of ilium |
| 80841 | Displaced avulsion fracture of left ilium, initial encounter for | Closed fracture of ilium |
| 80841 | closed fracture Displaced avulsion fracture of unspecified ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Nondisplaced avulsion fracture of right ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Nondisplaced avulsion fracture of left ilium, initial encounter | Closed fracture of ilium |
| 80841 | for closed fracture Nondisplaced avulsion fracture of unspecified ilium, initial | Closed fracture of ilium |
| 80841 | encounter for closed fracture Other fracture of right ilium, initial encounter for closed | Closed fracture of ilium |
| 80841 | fracture Other fracture of left ilium, initial encounter for closed | Closed fracture of ilium |
| | fracture | Closed fracture of ilium |
| | closed fracture | |
| | closed fracture | Closed fracture of ischium |
| | closed fracture | Closed fracture of ischium |
| 80842 | for closed fracture | Closed fracture of ischium |
| 80842 | Displaced avulsion fracture of left ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Displaced avulsion fracture of unspecified ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of right ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of left ischium, initial encounter for closed fracture | Closed fracture of ischium |
| 80842 | Nondisplaced avulsion fracture of unspecified ischium, initial | Closed fracture of ischium |
| 80842 | Other specified fracture of right ischium, initial encounter for | Closed fracture of ischium |
| 80842 | Other specified fracture of left ischium, initial encounter for | Closed fracture of ischium |
| 80842 | Other specified fracture of unspecified ischium, initial | Closed fracture of ischium |
| 80849 | Fracture of unspecified parts of lumbosacral spine and pelvis, | Closed fracture of other specified part of pelvis |
| 80851 | Unspecified fracture of right ilium, initial encounter for open | Open fracture of ilium |
| 80851 | Unspecified fracture of left ilium, initial encounter for open | Open fracture of ilium |
| 80851 | Displaced avulsion fracture of right ilium, initial encounter | Open fracture of ilium |
| | 8083<br>8083<br>8083<br>8083<br>8083<br>80841<br>80842 | open fracture 8083 Fracture of superior rim of unspecified pubis, initial encounter for open fracture 8083 Other specified fracture of right pubis, initial encounter for open fracture 8083 Other specified fracture of left pubis, initial encounter for open fracture 8083 Other specified fracture of unspecified pubis, initial encounter for open fracture 80841 Unspecified fracture of right ilium, initial encounter for closed fracture 80841 Unspecified fracture of left ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of left ilium, initial encounter for closed fracture 80841 Displaced avulsion fracture of unspecified ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of right ilium, initial encounter for closed fracture 80841 Nondisplaced avulsion fracture of unspecified ilium, initial encounter for closed fracture 80841 Other fracture of right ilium, initial encounter for closed fracture 80841 Other fracture of right ilium, initial encounter for closed fracture 80841 Other fracture of unspecified ilium, initial encounter for closed fracture 80842 Unspecified fracture of right ischium, initial encounter for closed fracture 80842 Unspecified fracture of right ischium, initial encounter for closed fracture 80842 Unspecified fracture of left ischium, initial encounter for closed fracture 80842 Displaced avulsion fracture of right ischium, initial encounter for closed fracture 80842 Displaced avulsion fracture of right ischium, initial encounter for closed fracture 80842 Other specified fracture of left ischium, initial encounter for closed fracture 80842 Nondisplaced avulsion fracture of unspecified ischium, initial encounter for closed fracture 80842 Other specified fracture of right ischium, initial encounter for closed fracture 80843 Unspecified fracture of |


| 82535 | Nondisplaced fracture of fourth metatarsal bone, unspecified | Open fracture of metatarsal bone(s) |
|---|---|---|
| 82535 | Displaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Displaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Displaced fracture of fifth metatarsal bone, unspecified foot, | Open fracture of metatarsal bone(s) |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, right foot, | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | · |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Unspecified physeal fracture of right metatarsal, initial | Open fracture of metatarsal bone(s) |
| 82535 | Unspecified physeal fracture of left metatarsal, initial | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type I physeal fracture of right metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | initial encounter for open fracture Salter-Harris Type I physeal fracture of left metatarsal, | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | |
| 82535 | Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type II physeal fracture of left metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type III physeal fracture of right metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type III physeal fracture of left metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | .,, |
| 82535 | Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Other physeal fracture of right metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Other physeal fracture of left metatarsal, initial encounter | Open fracture of metatarsal bone(s) |
| 82539 | Fracture of unspecified metatarsal bone(s), right foot, initial | Other open fracture of tarsal and metatarsal bones |
| 82539 | Fracture of unspecified metatarsal bone(s), left foot, initial | Other open fracture of tarsal and metatarsal bones |
| 8260 | encounter for open fracture Displaced unspecified fracture of right great toe, initial | Closed fracture of one or more phalanges of foot |
| 0260 | encounter for closed fracture | Classifications of any angular photographs |
| 8200 | encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced unspecified fracture of right great toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced unspecified fracture of left great toe, initial | Closed fracture of one or more phalanges of foot |
| 8260 | Displaced fracture of proximal phalanx of right great toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Displaced fracture of proximal phalanx of left great toe, | Closed fracture of one or more phalanges of foot |
| 8260 | initial encounter for closed fracture Displaced fracture of proximal phalanx of unspecified great | Closed fracture of one or more phalanges of foot |
| 0260 | toe, initial encounter for closed fracture | Closed fronting of any an array whelever a fifty |
| | initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced fracture of proximal phalanx of left great toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced fracture of proximal phalanx of unspecified | Closed fracture of one or more phalanges of foot |
| | 82535<br>82536<br>82536<br>82536<br>82536<br>82537<br>82539<br>8260 | foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Unspecified physeal fracture of right metatarsal, initial encounter for open fracture Septimental fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type I physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type III physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type III physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fract |


| | 1 | |
|---|---|---|
| 8260 | Other fracture of right lesser toe(s), initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Other fracture of left lesser toe(s), initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Other fracture of unspecified lesser toe(s), initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified fracture of right toe(s), initial encounter for | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified fracture of left toe(s), initial encounter for closed | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified fracture of unspecified toe(s), initial encounter for | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified physeal fracture of phalanx of right toe, initial | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified physeal fracture of phalanx of left toe, initial | Closed fracture of one or more phalanges of foot |
| 8260 | Unspecified physeal fracture of phalanx of unspecified toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type I physeal fracture of phalanx of right toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type I physeal fracture of phalanx of left toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type I physeal fracture of phalanx of unspecified | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type II physeal fracture of phalanx of right toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type II physeal fracture of phalanx of left toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type II physeal fracture of phalanx of | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type III physeal fracture of phalanx of right toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type III physeal fracture of phalanx of left toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type III physeal fracture of phalanx of | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type IV physeal fracture of phalanx of right toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type IV physeal fracture of phalanx of left toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Salter-Harris Type IV physeal fracture of phalanx of | Closed fracture of one or more phalanges of foot |
| 8260 | Other physeal fracture of phalanx of right toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Other physeal fracture of phalanx of left toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Other physeal fracture of phalanx of unspecified toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8261 | Displaced unspecified fracture of right great toe, initial | Open fracture of one or more phalanges of foot |
| 8261 | Displaced unspecified fracture of left great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| 8261 | Nondisplaced unspecified fracture of right great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| 8261 | Nondisplaced unspecified fracture of left great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| 8261 | Displaced fracture of proximal phalanx of right great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| 8261 | Displaced fracture of proximal phalanx of left great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| 8261 | Displaced fracture of proximal phalanx of unspecified great toe, initial encounter for open fracture | Open fracture of one or more phalanges of foot |
| | 8260 | dosed fracture 8260 Other fracture of left lesser toe(s), initial encounter for closed fracture 8260 Unspecified fracture of unspecified lesser toe(s), initial encounter for closed fracture 8260 Unspecified fracture of right toe(s), initial encounter for closed fracture 8260 Unspecified fracture of left toe(s), initial encounter for closed fracture 8260 Unspecified fracture of unspecified toe(s), initial encounter for closed fracture 8260 Unspecified physeal fracture of phalanx of right toe, initial encounter for closed fracture 8260 Unspecified physeal fracture of phalanx of left toe, initial encounter for closed fracture 8260 Unspecified physeal fracture of phalanx of unspecified toe, initial encounter for closed fracture 8260 Unspecified physeal fracture of phalanx of unspecified toe, initial encounter for closed fracture 8260 Salter-Harris Type I physeal fracture of phalanx of right toe, initial encounter for closed fracture 8260 Salter-Harris Type I physeal fracture of phalanx of unspecified toe, initial encounter for closed fracture 8260 Salter-Harris Type I physeal fracture of phalanx of right toe, initial encounter for closed fracture 8260 Salter-Harris Type II physeal fracture of phalanx of right toe, initial encounter for closed fracture 8260 Salter-Harris Type II physeal fracture of phalanx of left toe, initial encounter for closed fracture 8260 Salter-Harris Type III physeal fracture of phalanx of left toe, initial encounter for closed fracture 8260 Othe |


## Appendix A Frailty markers


## Falls


## Appendix A Frailty markers

### Combined Comorbidity Score for Claims Data

Gagne II, Glynn RI, Avorn I, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her O. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


## Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

### Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

### Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| And epiceptic non-mood stabilizers | |
|------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

#### Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

### Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

#### Selective serotonin reuptake inhibitor

| Total and the second se | |
|---|---|
| NDC Generic Name | |
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

### Tricyclic antidepressants

| NDC Generic Name | |
|------------------------------------|--------------------------------|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL |
| AMOXAPINE | DOXEPIN HCL |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL |

### Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

## Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM, PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM,PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM, PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| Antiplatelet agents | |
|---|---|
| NDC Generic Name | |
| ABCIXIMAB | CILOSTAZOL |
| ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | VORAPAXAR SULFATE |
| NDC Brand Name | |
| ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

## Angiotensin II Receptor Blockers

| NDC Generic Name | |
|---|---|
| ALISKIREN/VALSARTAN | LOSARTAN POTASSIUM |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE/VALSARTAN | OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZID |
| AZILSARTAN MEDOXOMIL | OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE | TELMISARTAN |
| CANDESARTAN CILEXETIL | TELMISARTAN/AMLODIPINE BESYLATE |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE | TELMISARTAN/HYDROCHLOROTHIAZIDE |
| IRBESARTAN | VALSARTAN |

| IRBESARTAN/HYDROCHLOROTHIAZIDE | VALSARTAN/HYDROCHLOROTHIAZIDE |
|--------------------------------|--------------------------------|
| NDC Brand Name | |
| AMLODIPINE-VALSARTAN | EXFORGE HCT |
| ATACAND | HYZAAR |
| ATACAND HCT | IRBESARTAN |
| AVALIDE | IRBESARTAN-HYDROCHLOROTHIAZIDE |
| AVAPRO | LOSARTAN POTASSIUM |
| AZOR | LOSARTAN-HYDROCHLOROTHIAZIDE |
| BENICAR | MICARDIS |
| BENICAR HCT | MICARDIS HCT |
| CANDESARTAN CILEXETIL | TELMISARTAN |
| CANDESARTAN-HYDROCHLOROTHIAZID | TELMISARTAN-AMLODIPINE |
| COZAAR | TELMISARTAN-HYDROCHLOROTHIAZID |
| DIOVAN | TRIBENZOR |
| DIOVAN HCT | TWYNSTA |
| EDARBI | VALSARTAN |
| EDARBYCLOR | VALSARTAN-HYDROCHLOROTHIAZIDE |
| EXFORGE | VALTURNA |

| Angiotensin Converting Enzyme inhibitors | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | LISINOPRIL |
| BENAZEPRIL HCL | LISINOPRIL/HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE | MOEXIPRIL HCL |
| CAPTOPRIL | MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | PERINDOPRIL ERBUMINE |
| ENALAPRIL MALEATE | QUINAPRIL HCL |
| ENALAPRIL MALEATE/FELODIPINE | QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE | RAMIPRIL |
| ENALAPRILAT DIHYDRATE | TRANDOLAPRIL |
| FOSINOPRIL SODIUM | TRANDOLAPRIL/VERAPAMIL HCL |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ACCUPRIL | LOTREL |
| ACCURETIC | LYTENSOPRIL |
| ACEON | LYTENSOPRIL-90 |
| ALTACE | MAVIK |
| AMLODIPINE BESYLATE-BENAZEPRIL | MOEXIPRIL HCL |
| BENAZEPRIL HCL | MOEXIPRIL-HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL-HCTZ | MONOPRIL |
| BENAZEPRIL-HYDROCHLOROTHIAZIDE | MONOPRIL HCT |
| CAPOTEN | PERINDOPRIL ERBUMINE |
| CAPOZIDE | PRINIVIL |
| CAPTOPRIL | PRINZIDE |
| CAPTOPRIL-HYDROCHLOROTHIAZIDE | QUINAPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | QUINAPRIL HCL |
| ENALAPRIL MALEATE | QUINAPRIL-HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE-HCTZ | QUINARETIC |
| ENALAPRIL MALEATE/HCTZ | RAMIPRIL |
| ENALAPRIL-HYDROCHLOROTHIAZIDE | TARKA |
| ENALAPRILAT | TRANDOLAPRIL |
| EPANED | TRANDOLAPRIL-VERAPAMIL |
| FOSINOPRIL SODIUM | UNIRETIC |
| FOSINOPRIL-HYDROCHLOROTHIAZIDE | UNIVASC |
| LEXXEL | VASERETIC |
| LISINOPRIL | VASOTEC |
| LISINOPRIL-HCTZ | VASOTEC I.V. |
| LISINOPRIL-HYDROCHLOROTHIAZIDE | ZESTORETIC |
| LOTENSIN | ZESTRIL |
| LOTENSIN HCT | |

### Beta blockers

| NDC Generic Name | |
|-------------------------|------------------------------------------|
| ACEBUTOLOL HCL | ESMOLOL HCL |
| ATENOLOL | LABETALOL HCL |
| ATENOLOL/CHLORTHALIDONE | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| BISOPROLOL FUMARATE | METOPROLOL TARTRATE |

| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE | METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
|---|---|
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE | NEBIVOLOL HCL |
| CARTEOLOL HCL | SOTALOL HCL |
| CARVEDILOL | TIMOLOL |
| CARVEDILOL PHOSPHATE | TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE | TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF | TIMOLOL MALEATE/PF |
| NDC Brand Name | |
| ACEBUTOLOL HCL | ISTALOL |
| ATENOLOL | KERLONE |
| ATENOLOL W/CHLORTHALIDONE | LABETALOL HCL |
| ATENOLOL-CHLORTHALIDONE | LOPRESSOR |
| BETAPACE | LOPRESSOR HCT |
| BETAPACE AF | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL TARTRATE |
| BETIMOL | METOPROLOL-HYDROCHLOROTHIAZIDE |
| BETOPTIC | NORMODYNE |
| BETOPTIC S | OCUPRESS |
| BISOPROLOL FUMARATE | SECTRAL |
| BISOPROLOL FUMARATE-HCTZ | SENORMIN |
| BISOPROLOL FUMARATE/HCTZ | SORINE |
| BISOPROLOL-HYDROCHLOROTHIAZIDE | SOTALOL |
| BLOCADREN | SOTALOL AF |
| BREVIBLOC | SOTALOL HCL |
| BYSTOLIC | TENORETIC 100 |
| CARTEOLOL HCL | TENORETIC 50 |
| CARTROL | TENORMIN |
| CARVEDILOL | TENORMIN CALENDAR PAK |
| COMBIGAN | TIMOLIDE |
| COREG | TIMOLOL MALEATE |
| COREG CR | TIMOPTIC |
| COSOPT | TIMOPTIC OCUDOSE |
| COSOPT PF | TIMOPTIC-XE |
| DORZOLAMIDE-TIMOLOL | TOPROL XL |
| DUTOPROL | TRANDATE |
| ESMOLOL HCL | ZEBETA |
| HYPERTENSOLOL | ZIAC |

### Calcium channel blockers

| Calcium channel blockers | |
|---|---|
| HCPCS | |
| C9248 | |
| NDC Generic Name | |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE | BEPRIDIL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE | CLEVIDIPINE BUTYRATE |
| AMLODIPINE BESYLATE | DILTIAZEM HCL |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | DILTIAZEM MALATE |
| AMLODIPINE BESYLATE/VALSARTAN | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |

| NYMALIZE |
|------------------------|
| PLENDIL |
| POSICOR |
| PROCARDIA |
| PROCARDIA XL |
| SULAR |
| TARKA |
| TAZTIA XT |
| TEKAMLO |
| TELMISARTAN-AMLODIPINE |
| TIAMATE |
| TIAZAC |
| TRANDOLAPRIL-VERAPAMIL |
| TRIBENZOR |
| TWYNSTA |
| VASCOR |
| VERAPAMIL ER |
| VERAPAMIL ER PM |
| VERAPAMIL HCL |
| VERAPAMIL SR |
| VERELAN |
| VERELAN PM |

### Diuretics

| NDC Generic Name | |
|-----------------------------------|---------------------|
| AMILORIDE HCL | HYDROCHLOROTHIAZIDE |
| AMILORIDE HCL/HYDROCHLOROTHIAZIDE | HYDROFLUMETHIAZIDE |
| BENDROFLUMETHIAZIDE | INDAPAMIDE |
| BUMETANIDE | METHYCLOTHIAZIDE |
| CHLOROTHIAZIDE | METOLAZONE |
| CHLORTHALIDONE | POLYTHIAZIDE |
| EPLERENONE | SPIRONOLACTONE |
| ETHACRYNATE SODIUM | TORSEMIDE |
| ETHACRYNIC ACID | TRIAMTERENE |
| FUROSEMIDE | TRICHLORMETHIAZIDE |

## Nitrates

| Nitrates | |
|---|---|
| NDC Generic Name | |
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL NITROGLYCERIN/DEXTROSE 5 % IN WATER | |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |
| DILATRATE-SR | NITROCINE |
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 NITROMIST | |
| OREX-2.5 NITRONAL | |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |

| ISOTRATE ER | NITROSTAT IV |
|--------------------------|-----------------|
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| Lipid lowering drugs | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | METHYLTETRAHYDROFOLATE GLUCOSAMINE/NIACINAMIDE/CUPRIC &ZN OX |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA | NIACIN |
| ATORVASTATIN CALCIUM | NIACIN (INOSITOL NIACINATE) |
| BETA-CAROTENE(A) W-C & E/NIACINAMIDE/VIT B2/LUT/MIN/GLU-ONE | NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| CERAMIDES 1,3,6-11/NIACINAMIDE | NIACIN/LOVASTATIN |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID | NIACIN/SIMVASTATIN |
| CHOLESTYRAMINE | NIACINAMIDE |
| CHOLESTYRAMINE (WITH SUGAR) | NIACINAMIDE ASCORBATE |
| CHOLESTYRAMINE/ASPARTAME | NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| COLESEVELAM HCL | NIACINAMIDE/RIBOFLAVIN/BETA-CAROTENE(A) W-C & E/MINERALS |
| COLESTIPOL HCL | NIACINAMIDE/VIT B6/VIT C/FA/COPPER/MG CIT/ZN GLUC/ALIP ACID |
| EZETIMIBE | PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| EZETIMIBE/ATORVASTATIN CALCIUM | PITAVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN | POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| FENOFIBRATE | PRAVASTATIN SODIUM |
| FENOFIBRATE NANOCRYSTALLIZED | ROSUVASTATIN CALCIUM |
| FENOFIBRATE,MICRONIZED | SIMVASTATIN |
| FLUVASTATIN SODIUM | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| FOLIC ACID/NIACINAMIDE/ZINC | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| GEMFIBROZIL | THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| INOSITOL NIACINATE | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |

### Non-insulin diabetes medications

| NOT-HISUITI GIADETES THEGICATIONS | |
|---|---|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL PIOGLITAZONE HCL/METFORMIN HCL | |
| CANAGLIFLOZIN/METFORMIN HCL REPAGLINIDE | |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |

| GLYBURDE/METFORMIN HCL UNAGUPTIN METFORNININ ACARDOSE LCN-TOLAM ACACTOHLUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTORIS JANUMET XR JANUMET XR JANUMET XR AMARYL JANUVIA APPFORNININ JENITADULETO APPEORNININ JENITADULETO APPEORNININ JENITADULETO AVANDAMET A | GLYBURIDE | SAXAGLIPTIN HCL |
|---|---|---|
| INAGIPTIN/METFORMIN HCI. METFORMIN HCI. METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOUNE METFORMIN/CAFFEIRE/AMINO ACIDS #7/HERBAL COMB.#125/CHOUNE BIT TOLBUTAMIDE METFORMIN/CAFFEIRE/AMINO ACIDS #7/HERBAL COMB.#125/CHOUNE BIT TOLBUTAMIDE MOD Brand Name ACARBOSE ACATOPLUS MET ACTOPLUS MET ACTOPLUS MET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTORIUS MET INVOKAMET A | GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| METFORMIN HCL METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE METFORMIN/CAFFEINE/AMINO ACIDS.#7/HERBAL COMB.#125/CHOLINE METFORMIN/CAFFEINE/AMINO ACIDS.#7/HERBAL COMB.#125/CHOLINE BIT MDC Brand Name ACARBOSE ICN-TOLAM ACACROSE ICN-TOLAM ACTOPLUS MET ACTOPLUS MET ACTOPLUS MET INVOKAMET ACTOS JANUMET INVOKAMET APPFORNIND JUVISYNC AVANDAMET AVANDAMET AVANDAMET AVANDAWI AVANDAWI AVANDAWI CHLORABETIC 250 METFORMIN HCL CHLORABETIC 250 METFORMIN HCL ER DIABIESE DIABIESE DIABIESE DIABIESE DIABIESE NATEGLINDE DIBABTAO DUSTACT ONGLYZA DYMELOR FORTAMET ORINASE GLIMEPRIDE GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KR GLIUCOPHAGE PRECOSE GLIUCOPHAGE | LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB#125/CHOUNE BIT NDC Brand Name ACARBOSE ICN-TOLBUT MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET NI ANUMET NI ACTORIUS MET NI ANUMET NI ANUMET NI ACTORIUS MET NI APPEORMIN IENTADUETO IPUTISTNC AVANDARY AVANDARY AVANDARY AVANDIA CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 ACTORIUS METFORMIN HCL CHURRABETIC 250 CHURLABETIC MICRONASE DIBBITIC ONGLYZA | LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| MDC Brand Name ACARBOSE ACETOHEXAMIDE ACAROSE ICN-TOLAM ACETOHEXAMIDE INSULASE ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET (ACTORIUS MET ( | METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| MDC Brand Name ACARBOSE ACETOHEXAMIDE ACAROSE ICN-TOLAM ACETOHEXAMIDE INSULASE ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET (ACTORIUS MET ( | METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | TOLAZAMIDE |
| ACARBOSE ACTOPLUS MET INSULASE INSULASE ACTOPLUS MET XR ACTOPLUS MET XR JANUMET XR ACTOPLUS MET XR JANUMET XR ACTOPLUS MET XR JANUMET XR AMARYL APPEORMIN JENITADUETO JUVISYNC AVANDAMET KAZANO AVANDIA CHLORABETIC 250 METFORMIN HCL METFORMIN HCL CHLORABETIC 250 METFORMIN HCL | | TOLBUTAMIDE |
| ACTOPLUS MET INVOKAMET ACTOPUS MET XR ACTOPUS MET XR JANUMET ACTOS JANUMET ACTOS JANUMET XR ACTOPUS MET XR ACTOPUS MET XR ACTOS JANUMET XR AMARYL APPFORMIN JENTADUETO APPFORMINO JUVISYNC APANDAMET KAZANO AVANDAMET KAZANO AVANDAMET ACTOR AVANDAMET AVANDAMET AVANDAMET ACTOR AVANDAMET AVANDAMET AVA | NDC Brand Name | |
| ACTOPLUS MET XR JANUMET ACTOPUS MET XR JANUMET R ACTOS JANUMET XR AMARYL JANUVIA APPFORMIN JANUVIA APPFORMIND JUVISYNC AVANDAMET KAZANO AVANDAMET KAZANO AVANDAMYL KOMBIGLYZE XR AVANDIA METFORMIN HCL CHLORABETIC 250 M | ACARBOSE | ICN-TOLAM |
| ACTOPLUS MET XR ACTOS JANUMET ACTOS JANUMET XR AMARYL APPFORMIN APPFORMIN JENTADUETO APPFORMIN-D JUVISYNC KAZANO AVANDAMET KAZANO AVANDAMET AVANDARYL AVANDARYL KOMBIGLYZE XR AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORAPROPAMIDE MICRONASE DIABITESE NATEGLINDE JIBAITROL DIBAITROL DIBATROL DIBATROL DIBATROL DIBATROL DIBATROL ORNETIC GUNPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE RR GUIPZIDE XL GUIPZIDE KR GUIPZIDE METFORMIN GUILAZONE-GUIMEPRIDE GUIPZIDE KR GUIPZIDE METFORMIN GUILAZONE-GUIMEPRIDE GUIPZIDE METFORMIN GUILAZONE-GUIMEPRIDE GUIPZIDE METFORMIN GUILAZONE-GUIMEPRIDE GUIPZIDE-METFORMIN GUILAZONE-GUIMEPRIDE GUIDAZONE-GUIMEPRIDE GUIDAZO | ACETOHEXAMIDE | INSULASE |
| ACTOS JANUMET XR AMARYL JANUVIA APPEORMIN APPEORMIN APPEORMIND APPEORMIND APPEORMIND AVANDAMET KAZANO AVANDAMET KAZANO AVANDARYL KOMBIGIYZE XR AVANDIA CHLORABETIC 250 METFORMIN HCL CHLORRPROPAMIDE METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABITASE NATEGUNIDE DIBABTA NESINA DIABITACI NESINA DUETACT ONGIYZA DYMELOR FORTAMET ORINASE GUMEPIRIDE OSENI GUIPZIDE GUIPZIDE X GUIPZIDE X GUIPZIDE AMETFORMIN GULCAMIDE GUIPZIDE METFORMIN GULCAMIDE GUIPZIDE METFORMIN GULCAMIDE GUICAMIDE GUICAMIDE GUICAMIDE GUICAMIDE FORDAMET GUICAMIDE GUIVBURIDE GUICAMIDE GUIVBURIDE | ACTOPLUS MET | INVOKAMET |
| AMARYL APPFORMIN JENTADUETO APPFORMIN-D JUVISYNC AVANDAMET KAZANO AVANDARYT KOMBIGLYZE XR AVANDIA WETAGUP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE MICROMASE DIABITA DIBATROL DIBATROL DIBATROL DIBATROL ONGIYZA DYMELOR FORTAMET GUILPIZIDE GUIPZIDE ER GUIPZIDE ER PIOGLITAZONE-GUIMEPIRIDE GUIPZIDE XL GUIPZIDE XL GUIPZIDE METFORMIN GULCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOTROL KL GUINETA STARIK GLUCOTROL KL GUINETA GLUCOTROL KL GUINETA GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOPHAGE GLUCOPHA | ACTOPLUS MET XR | JANUMET |
| APPFORMIND APPFORMIND APPFORMIND APPFORMIND AVANDAMET KAZANO AVANDAMET KAZANO AVANDARYL KOMBIGLYZE XR AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABITA MICRONASE DIABITA MICRONASE DIBAITAOL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET GUIMEPIRIDE GUIPZIDE PIOGUITAZONE HCL GUIPZIDE ER GUIPZIDE RT GUIPZIDE AUTORIA PRANDINE GUIPZIDE-METFORMIN PRANDIMET GUICOPHAGE PRECOSE GUICOPHAGE PRECOSE GUICOPHAGE GUICOTROL XL ROMASE GUIMETIA GUICOVANCE SK-TOLBUTADE GUIVERIDE GUINETOR GUINETOR GUINETOR GUINETOR GUINETOR GUINETOR GUINETOR GUICOTROL XL ROMASE GUINETOR GUINETOR GUINETOR GUICOVANCE SK-TOLBUTADOR GUIVASE GUIVASE FRANDIN GUIVASE FRANDIR GUIVASE FRANDIR GUIVANDE GUIVASE FRANDIR GUICOVANCE GUIVERIDE GUIVASE FRANDIR GUIVANSE FRANDIR GUIVASE | ACTOS | JANUMET XR |
| APPFORMIN-D AVANDAMET KAZANO AVANDAMET KAZANO AVANDAYL KOMBIGIVZE XR AVANDIA CHIORABETIC 250 METFORMIN HCL CHIORABETIC 250 METFORMIN HCL ER DIABETA MICRONASE DIABIRSE MATEGINIDE DIBATROL DUETACT ONGLYZA DYMELOR OFFICE GUIPZIDE GUIPZIDE GUIPZIDE XL GUIPZIDE XL GUIPZIDE XL GUIPZIDE XL GUIPZIDE METFORMIN GUICOTROL GUIPZIDE MICRONIZED GUIPZIDE MICRONIZED GUIVANDE GUIPZIDE MICRONIZED GUIPZIDE MICRONIZED GUIVANDE GUIPZIDE MICRONIZED GUIPZIAMIDE GUIP | AMARYL | JANUVIA |
| AVANDAMET AVANDARYL KAZANO KAZANO KAYANDIA METAGUP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABIESA MICRONASE DIABINESE NATEGUNIDE DIBATROL DUFFACT ONGLYZA DYMELOR FORTAMET GUMEPRIDE GUPZIDE ER GUPZIDE ER GUPZIDE ER GUINZIDE AUGUNDE GULCOPHAGE GLUCOPHAGE GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLUCO | APPFORMIN | JENTADUETO |
| AVANDIAYL AVANDIA AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL DUETACT ONGLYZA DYMELOR ORINASE GLIPIZIDE GLIPIZIDE GLIPIZIDE GLIPIZIDE R GLIPIZIDE XL GLIPIZ | APPFORMIN-D | JUVISYNC |
| AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL NESINA DUFTACT ONGLYZA DYMELOR ORIBETIC GUIMEPRIDE GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE NETFORMIN PRANDIMET GLUCOPHAGE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPORTED GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYNASE TOLAMIDE GLYNASE TRADJETNAMI GLYNASE GLYNASE TRADJETNAMI GLYCONICA GRACE GRACH GRACH GLYCONICA GRACH GLYCONICA GLYCONICA GLYCONICA GLYCONICA GLYCONICA GLYCONICA GRACH GLYCONICA GLYCONICA GRACH GLYCONICA GLYCONICA GLYCONICA GRACH GLYCONICA GRACH GRACH GLYCONICA GRACH GLYCONICA GLYCONICA GRACH | AVANDAMET | KAZANO |
| CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL NESINA DUETACT ONGLYZA DYMELOR FORTAMET ORINASE GLIMEPIRIDE GLIPIZIDE GLIPIZIDE R GLIPIZIDE R GLIPIZIDE XL GLIPIZIDE XL GLIPIZIDE METFORMIN GLICAMIDE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOTROL GLUCOTROL GLICOTROL G | AVANDARYL | KOMBIGLYZE XR |
| CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE NATEGLINIDE DIBATROL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC GUMEPRIDE OSENI GUIPIZIDE R GUIPIZIDE R GUIPIZIDE R GUIPIZIDE XL GUIPIZIDE XL GUIPIZIDE XL GUIPIZIDE XL GUIPIZIDE METFORMIN GUICOPHAGE GUICOPHAGE GUICOPHAGE GUICOPHAGE GUICOPHAGE GUICOTROL GUICOTROL GUICOTROL GUICOPHACE | AVANDIA | METAGLIP |
| DIABETA MICRONASE DIABNIESE NATEGLINIDE DIBATROL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE RIPIZIDE PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIME GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLBUTAMISE GLYCON GLYCON GLYCON GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON TOLBUTAMIDE GLYCON GRACH | CHLORABETIC 250 | METFORMIN HCL |
| DIABINESE DIBATROL DIBATROL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE GIPIZIDE R GIPIZIDE R GIPIZIDE R GUIPIZIDE R GUICONAGE GUIPIZIDE R GRANDIN GRANDIMET GLUCAMIDE FRANDIME GLUCOPHAGE PRANDIN GLUCOPHAGE REPAGLINIDE GLUCOPHAGE R GUCOPHAGE R GUCOPHAGE R GUCOYNOL RIOMET GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLINASE GLYCON GLYNASE TRADJENTA | CHLORPROPAMIDE | METFORMIN HCL ER |
| DIBATROL DUETACT DUETACT DOMGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE R PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCOPHAGE PRANDIN GLUCOPHAGE RUCOPHAGE RUCOPHAGE RUCOTROL RUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL ROMASE GLUCOTROL ROMASE GLUCOTROL GLUCOTROL GLUCOTROL SCHOOL GLUCOTROL GLUCOTRO | DIABETA | MICRONASE |
| DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GUPIZIDE PIOGLITAZONE HCL GUPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLBUTAMIDE GLYCON TOLINASE GLYNASE TRADJENTA | DIABINESE | NATEGLINIDE |
| DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE RIPIGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN GLIPIZIDE-METFORMIN GLICOPHAGE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL GLUCOTROL GLUCOTROL RIOMET GLUCOVANCE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE | DIBATROL | NESINA |
| FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIME GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLUMETZA STARLIX GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLBUTAMIDE GLYCRON TOLBUTAMIDE GLYCRON TOLBUTAMIDE GLYCRON TOLINASE GLYCRON TOLINASE GLYCRON TOLINASE | DUETACT | ONGLYZA |
| GLIMEPIRIDE GLIPIZIDE GLIPIZIDE GLIPIZIDE ER GLIPIZIDE ER GLIPIZIDE XL PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLYBURIDE GLY | DYMELOR | ORIBETIC |
| GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | FORTAMET | ORINASE |
| GLIPIZIDE ER GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLUCOVANCE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYCRON TOLBUTAMIDE GLYBURIDE GLYBURI | GLIMEPIRIDE | OSENI |
| GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL ROMASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES | GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE-METFORMIN GLUCAMIDE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE PRECOSE GLUCOPHAGE XR GLUCOTROL GLUCOTROL GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE G | GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL ROMASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES GLYBURIDE TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES GLYBURIDES GLYNASE TRADJENTA | GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLUCOPHAGE PRECOSE GLUCOPHAGE XR REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYRON TOLINASE GLYNASE TRADJENTA | GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCOPHAGE XR GLUCOTROL GLUCOTROL XL GLUCOTROL XL RONASE GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCAMIDE | PRANDIN |
| GLUCOTROL GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE GLYBURIDE GLYBURIDE TOLAMIDE GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOPHAGE | PRECOSE |
| GLUCOTROL XL GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOTROL | RIOMET |
| GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOTROL XL | RONASE |
| GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOVANCE | SK-TOLBUTAMIDE |
| GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUMETZA | STARLIX |
| GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE | TOLAMIDE |
| GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| | GLYCRON | TOLINASE |
| GLYSFT | GLYNASE | TRADJENTA |
| OLIGET | GLYSET | |

## Insulin


| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
|-----------------------------|--------------------------------|
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| HUMALOG MIX 50/50 | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | |

### Antidepressants

| HCPCS | |
|---|---|
| J1320 | |
| NDC Generic Name | |
| | IN ALDRA A ALAUS LLCI |
| AMITRIPTYLINE HCL IMIPRAMINE HCL | |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEVOMILNACIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT, MISC. COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE VORTIOXETINE HYDROBROMIDE | |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |

| AMONAPINE MINTAZAPHE ANYDROUS ANAPETAMIN PREDITAMONE PREDITAMONE NOFERAMIN NEFACOONE HCI NOFERAMIN NEFACOONE HCI NOFERAMIN NOFERAMIN NOFERAMIN NOFERAMIN NORTRIPTYLIN HCI OLANZARIMA HCI OLANZARIMA HCI SENDERIMA SENDER PAMELOR BUDEPRION SR BUDEPRION SR BUDEPRION SR PAMELOR BUDEPRION SR PARIC CR BUDEPRION MCI PARIC CR BUDEPRION MCI PARIC CR BUDEPRION MCI PERTIND BUDEPRION HCI PERTIND PERTIND BUDEPRION HCI PERTIND BUDEPRION HCI PERTIND BUDEPRION HCI PERTIND BUDEPRION HCI PERTIND PERTIND BUDEPRION HCI BUDEPRION HCI PERTIND BUDEPRION HCI BUDEPRION | AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
|---|---|---|
| AMAFABIL APRIEZIM NARONE APPRITAMONE NOBERAMI NO | · | |
| NEFACOONE INC. | | |
| MORFRANII | | |
| APSENDIN MORTAMINE HU. APSENDIN MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO MORTAMINE HU. AVENITY HU. BRIDDERICO M. BR | | |
| ASENDIN | | |
| AVENTYL HCL OLANAZARIK-FLUXXETINE HCL BRISTELIX BRISTELIX BRISTELIX DEFPROR N. BRISTELIX PARKICR BLUDEPRON X. PEXEVA PEXEVA PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. BLUPROPHON X. PEXEVA PROSE BLUPROPHON X. BLUPROPHON X. PROSE BLUPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. PROSE BLUPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUDEPROPHON X. BLUD X. BLUDEPROPHON X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDREPROM X. BLUDR | | |
| SINTELLIX OLEFTO & R | | |
| RRISDELLE PAMELOR PARCETINE H.C. PERPERBAN PARCETINE H.C. PERPERBAN PERPENBAN PERPENBA | | |
| BRUDEPRION SR | | |
| PAXIL PAXI | | |
| BURDEDAN PAXIL CR | | |
| BURDOPION H.C. PERTER | | |
| BURDOPION HCL ER BURDOPION HCL SR BURDOPION SC PEXEVA BURDOPION SC PEXEVA BURDOPION SC PERCENA PRISTIQ ER BURDOPION SC PROTECT | | |
| BURDOPION HCL SR | | |
| PURPOPION XL | | |
| CELEXA PROTREPTYLINE HCL CHTALOPRAM PROZAC CITALOPRAM HRR PROZAC REHIVE DESIPRAM DESVENILATANIE FROM DESVENILATANIE SERTRALINE HCL TRAVIL 10-2 | | |
| CHIORDIAZEPOXIDE-AMITRIPTYUNE PROZAC CITALOPRAM PROZAC CWERKLY PRUDOXIN CYMBALTA Q.E. L DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RAPIFLUX DECONIL RE-LUVE DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FU DESVENLAFAXINE FUMARATE ER SARAFEM SELFEMRA DOKERIH HCL SENTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE DOLOXETINE HCL SERTROXATINE PROLOXE PVILL 10 SERZONE PVILL 25 SINEQUAN SK-PAMITRIPTYUNE SK-PAMITRIPTY | | |
| CITALOPRAM HBR PROZAC C TITALOPRAM HBR PROZAC WEEKLY CICMIPPAMINE HCL PRUDOWN CYMBALTA Q.E.L PRUDOWN CICMIPPAMINE HCL PRUDOWN CESTINAL Q.E.L PRUDOWN DESIPHARMINE HCL RAPPILUX DESIPHARMINE HCL REHVE DESIPHARMINE HCL REHVE DESIVENLARAKINE ER REMERON DESVENLARAKINE ER SARAFEM DESVENLARAKINE FUMARATE ER SARAFEM DOXEPIN HCL SENTROXATINE DULOXEINIE HCL SENTROXATINE DULOXEINIE HCL SERTRALINE SERTRALINE SERTR | | |
| PROZAC WEEKLY | | |
| PRIDOXIN | | |
| CYMBALTA | | |
| DECONIL RAPIFLUX DESSIPRAMINE HCL RE-UVE DESSIPRAMINE HCL RE-UVE REMERON DESSIPRAMINE FUNARATE ER REMERON DESSURLAFAXINE FUMARATE ER SELFEMRA DOXEDIH HCL SERTROWATINE DOULOXETINE HCL SERTROWATINE SELFEMRA SILENOR E-VILL 100 SILENOR E-VILL 100 SILENOR E-VILL 55 SINEQUAN SERVALISO SK-AMITIRIPTYLINE E-VILL 50 SK-AMITIRIPTYLINE E-VILL 75 SK-PAMINE STABANIL STEFEXOR STABANIL SURMONTIL E-FEXOR SURMONTIL E-BAYL SURMONTIL E-MITRIP TOFRANIL-PM FINOVIL SYMBYAX SURMONTIL E-MITRIP TOFRANIL-PM FINOVIL TRAZAMINE E-SOTTALOPRAM OXALATE TRAZODONE HCL E-TRAFON 2-10 TRIAVIL 1-0 E-TRAFON 2-10 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 1-0 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-10 TRIAVIL 1-10 | | |
| DESIPRAMINE HCL DESVENLAFAXINE FUMARATE ER DESVENLAFAXINE MCL DULOXETINE HCL SERTROLATINE SERTROLATINE SERTROLATION SERTROLATINE SERTROLATION | | · · |
| DESVENLAFAXINE ER DESVENLAFAXINE FUMARATE ER DESYREL SELFEMRA DOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SERTRALINE SIMEQUAN SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SERTRALINE SOUTH TOFARAIL FINAPIL ENOPTH ENOPTH SERTRALINE SECTIALOPRAM OXALATE TRAZODONE HCL TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-10 TRANIL 2-5 TRANIL 2-6 TRANIL 2-7 TRANIL 2-7 TRANIL 2-8 TRANIL 2-9 TRANIL 2-9 TRANIL 2-10 TRANIL 2-1 | | |
| DESVENLAFAXINE FUMARATE ER SERFEMRA DOSYPRIL SELFWRA DOSYPRIL SELFWRA DOLOXEPIN HCL SENTROXATINE DULOXETINE HCL SERTRALINE SIMEOUAN SERTRALINE SERTRALI | | |
| DESYREL DESYREL DESYREL DESPIRACATINE DOXEPIN HCL SENTROXATINE DUICNETINE HCL SENTROXATINE DUICNETINE HCL SERZONE E-VILL 100 SIRNOR E-VILL 25 SINEQUAN SEVILL 25 SINEQUAN SK-RAMITRIPTYLINE E-VILL 50 SK-RAMITRIPTYLINE E-VILL 57 SK-PRAMINE STABANIL STABANIL STABANIL STABANIL SEFEXOR STABANIL SEMMONTIL ELAVIL SYMBYAX EMITRIP TOFRANIL FINDEP TOFRANILPM FINOVIL TRAZAMINE SECTIALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRAVIL 2-10 ETRAFON 2-10 TRAVIL 2-10 ETRAFON 2-10 TRAVIL 2-10 ETRAFON 4-10 TRAVIL 2-10 ETRAFON 4-10 TRAVIL 2-10 ETRAFON A-10 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON TORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON FORTE 4-25 TRAVIL 2-10 ETRAFON BORTE 4-25 TRAVIL 2-20 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-25 TRAVIL 2-3 ETRAFON BORTE 4-3 TRAVIL 2-3 ETRAFON BORTE 4-3 TRAVIL 2-3 ETRAFON BORTE 4-3 TRAVIL 2-3 TRAVIL 2-3 ETRAFON BORTE 4-3 TRAVIL 2-10 ETRAFON BORTE 4-3 TRAVIL 2-10 ETRAFON BORTE 4-3 E | | |
| DOUCRPIN HCL SERTRALINE HCL SILENOR SILENOR SILENOR SILENOR SILENOR SEAMITRIPTYLINE EVILL 75 SEPRAMINE SEFEXOR STABANIL SEFEXOR STABANIL SUMMONTIL SELAVIL SYMBYAX SILENOR SILENOR STABANIL SYMBYAX SILENOR STABANIL SELAVIL SELAVIL SELAV | | |
| DULOXETINE HCL SERTABLINE HCL SERZONE E-VILL 10 SERZONE E-VILL 25 SINEQUAN SILENOR E-VILL 25 SINEQUAN SINEQUAN SEPERSOR SEPERSOR STABANIL SEFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX SUMMONTIL LAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 2-10 TETRAFON 2-25 TRIAVIL 2-25 ETRAFON 2-10 TRIAVIL 2-25 ETRAFON 4-10 TRIAVIL 2-25 ETRAFON 1-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 ETRAFON FORTE 4-25 TRIAVIL 2-7 TRIAVIL 2-8 ETRAFON FORTE 4-25 TRIAVIL 2-9 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-26 ETRAFON FORTE 4-25 TRIAVIL 2-30 TRIAVIL 2-4 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-10 TRIAVI | | |
| E-VILL 10 SERZONE E-VILL 100 SILENOR E-VILL 25 SINEQUAN E-VILL 50 SK-AMITRIPTYLINE E-VILL 75 SK-PRAMINE EFFEKOR STABANIL EFFEKOR STABANIL EFFEKOR XR SURMONTIL LAVIL SYMBYAX EMITIRP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNAFOR 2-10 TRIAVIL 2-10 ETRAFON 3-10 TRIAVIL 2-10 ETRAFON 3-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 4-10 TRIAVIL 2-10 ETRAFON 1-10 TRIAVIL 2-10 | | |
| E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 25 SINEQUAN E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR STABANIL ELAVIL SYMBYAX EMITRIP ELAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL ENCOPLE ENCOPL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-10 ETRAFON 6-10 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 ETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON FORTE 4-25 FETRAFON TRIAVIL 5-4 FETRAFON TRIAVIL 5-5 FETRAFON TRIAVIL 5- | | |
| SINEQUAN | | |
| E-VILL 50 E-VILL 75 SK-PRAMINE EFFEXOR STABANIL EFFEXOR STABANIL EFFEXOR SYMBYAX ELAVIL SYMBYAX ELAVIL ELAVIL SYMBYAX ENTIFIP TOFRANIL-PM ENOUTH ENOUTH ENOUTH ENOUTH ENOUTH ETRACODONE HCL ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON BORTH 4-25 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2 | | |
| SK-PRAMINE | | |
| EFFEXOR STABANIL EFFEXOR XR SURMONTIL ELAVIL SYMBYAX EMITRP TOFRANIL ENDEP TOFRANIL-PM ENOVIL TRAZAMINE ENOVIL TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-5 ETRAFON 2-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 EFETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-10 FLUOX | | |
| SURMONTIL | | |
| ELAVIL SYMBYAX EMITRIP TOFRANIL ENDEP TOFRANIL ENDEP TOFRANIL-PM ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-5 ETRAFON 4-10 TRIAVIL 25-2 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-50 FLUOXETINE HCL TRIAVIL 4-50 FLUOXAMINE MALEATE TRIAVIL 4-50 FLUOXAMINE MALEATE TRIAVIL 4-50 FORFIVO XL VENLAFAXINE HCL EMANATE VIIBRYD EMINAVATE VIIBRYD EMINAVATE VIIBRYD EMINAVATE VIIBRYD EMINAMINE PAMOATE EMINAMINE PAMOATE EMINAMINE WELLBUTRIN SR EKENVIL WELLBUTRIN SR | | |
| EMITRIP ENDEP TOFRANIL ENDEP TOFRANILPM ENOVIL ENOVIL ENOVIL ETRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 TRIAVIL 2-5-2 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-50 FLUOVAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLOVOXAMINE MALEATE FLOVATE FORFIVO XL SABOXETINE VENLAFAXINE HCL MINAVATE | | |
| ENDEP FINDER FINDER FINOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETRAFON 2-10 TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 2-3 ETRIAVIL 2-40 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-5 ETRIAVIL 2-6 ETRIAVIL 2-7 ETRIAVIL 2-8 ETRIAVIL 3-9 ETRIAVIL | | STIVIDIAX |
| ENOVIL TRAZAMINE ESCITALOPRAM OXALATE TRAZODONE HCL ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 2-25 ETRAFON FORTE 4-25 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIAVIL 4-50 FUNDOXAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE MALEATE TRIMIPRAMINE HCL TRIAVIL 4-50 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL 25-5 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-50 TRIAVIL 2-5 TR | I E MITDID | TOFRANII |
| TRAZODONE HCL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 TRIAVIL 2-5 ETRAFON FORTE 4-25 TRIAVIL 2-6 FETZIMA TRIAVIL 2-7 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FORFIVO XL GABOXETINE GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL ER WANATE MIPPRAMINE HCL WINACTIL MIPRAMINE PAMOATE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-10 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2-5 TRIAVIL 2 | EMITRIP | |
| ETNOFRIL TRIAVIL 10-2 ETRAFON 2-10 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-2 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-10 FLUOXETINE HCL TRIAVIL 4-50 FLUOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FURD YENLAFAXINE HCL GABOXETINE WENLAFAXINE HCL WENLAFAXINE HCL ER WANATE WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WIBRYD WINFRAMINE HCL WINFRAMINE HCL WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT ZONALON | ENDEP | TOFRANIL-PM |
| ETRAFON 2-10 TRIAVIL 2-10 ETRAFON 2-25 TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FULOXETINE DR TRIAVIL 4-25 FULOXETINE HCL TRIAVIL 4-50 FULVOXAMINE MALEATE TRIMIPRAMINE MALEATE FULVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER IMIPRAMINE HCL VIVACTIL IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELBUTRIN JANIMINE WELBUTRIN SR KENVIL WELBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP<br>ENOVIL | TOFRANIL-PM<br>TRAZAMINE |
| TRIAVIL 2-25 ETRAFON A 4-10 TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUOXEMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FORFIVO XL VENLAFAXINE HCL VENLAFAXINE HCL MIPPAMINE HCL WIBRYD MIPPAMINE HCL WIBRYD WIBRYD MIPPAMINE HCL WINACTIL MIPPAMINE PAMOATE VELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO TRIAVIL 2-25 TRIAVIL 2-25 TRIAVIL 25-4 TRIAVIL 25-2 TRIAVIL | ENDEP ENOVIL ESCITALOPRAM OXALATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL |
| TRIAVIL 25-2 ETRAFON FORTE 4-25 TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMPRAMINE MALEATE TRIMPRAMINE MALEATE FORFIVO XL GABOXETINE WENLAFAXINE HCL WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WINAVATE WELBUTRIN JANIMINE JANIMINE KENVIL KHEDEZLA ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 |
| TRIAVIL 25-4 FETZIMA TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE HCL FLUVOXAMINE H | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 |
| TRIAVIL 4-10 FLUOXETINE DR TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 |
| TRIAVIL 4-25 FLUOXETINE HCL TRIAVIL 4-50 FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIBRYD VIMIPRAMINE HCL VIVACTIL VIVACTIL VIMIPRAMINE PAMOATE VELLBUTRIN VELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 |
| FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE WENLAFAXINE HCL VENLAFAXINE HCL ER WIBRYD WIBRYD WIBRYD WIBRYD WIMIPRAMINE HCL WINACTIL WIMIPRAMINE PAMOATE WELLBUTRIN JANIMINE KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 |
| TRIMIPRAMINE MALEATE FLUVOXAMINE MALEATE ER FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL VENLAFAXINE HCL GABOXETINE VENLAFAXINE HCL ER VIIBRYD VIIBRYD VIIBRYD VIIBRYD VIVACTIL | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 |
| FLUVOXAMINE MALEATE ER VANATRIP FORFIVO XL GABOXETINE VENLAFAXINE HCL ER VIBRYD VIBRYD VIVACTIL MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE VELBUTRIN VELBUTRIN SR KENVIL KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 |
| FORFIVO XL GABOXETINE WENLAFAXINE HCL ER WAVATE WIBRYD WIFRAMINE HCL WIFRAMINE HCL WIFRAMINE PAMOATE WELLBUTRIN WELLBUTRIN SR KENVIL KHEDEZLA KHEDEZLA ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 |
| GABOXETINE VENLAFAXINE HCL ER VIIBRYD IMIPRAMINE HCL VIVACTIL IMIPRAMINE PAMOATE WELLBUTRIN IANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VONLAFAXINE HCL ER VIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE |
| MAVATE VIBRYD MIPRAMINE HCL VIVACTIL MIPRAMINE PAMOATE WELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL KHEDEZLA ZOLOFT LEXAPRO VIBRYD VIVACTIL VEILBUTRIN SR WELLBUTRIN SL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP |
| MIPRAMINE HCL MIPRAMINE PAMOATE MELLBUTRIN JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO VIVACTIL WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL |
| IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER |
| JANIMINE WELLBUTRIN SR KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD |
| KENVIL WELLBUTRIN XL KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL |
| KHEDEZLA ZOLOFT LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN |
| LEXAPRO ZONALON | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL |
| LIMBITROL ZYBAN | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT |
| | ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA LEXAPRO | TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR WELLBUTRIN XL ZOLOFT ZONALON |

## Appendix A Comorbid conditions

**Atrial Fibrillation** 


## Appendix A Comorbid conditions


Heart Failure


| Dilation of Loft Padial Artory with Drug cluting Intraluminal | |
|---|---|
| , | |
| , | |
| Intraluminal Devices, Open Approach | |
| Dilation of Left Radial Artery with Four or More Drug- | |
| Intraluminal Devices, Open Approach | |
| Dilation of Left Radial Artery, Bifurcation, with Intraluminal | |
| Device, Open Approach– | |
| Dilation of Left Radial Artery with Intraluminal Device, Open | |
| Approach– | |
| Dilation of Left Radial Artery, Bifurcation, with Two | |
| Intraluminal Devices, Open Approach— | |
| Dilation of Left Radial Artery with Two Intraluminal Devices, | |
| Open Approach | |
| Dilation of Left Radial Artery, Bifurcation, with Three | |
| Intraluminal Devices, Open Approach– | |
| Dilation of Left Radial Artery with Three Intraluminal | |
| • | |
| Dilation of Left Radial Artery, Bifurcation, with Four or More | |
| • | |
| , | |
| 1 11 | |
| Intraluminal Device, Percutaneous Approach | |
| Dilation of Left Radial Artery with Drug-eluting Intraluminal | |
| Device, Percutaneous Approach-eluting Intraluminal Device, | |
| Percutaneous Approach | |
| Dilation of Left Radial Artery, Bifurcation, with Two Drug- | |
| eluting Intraluminal Devices, Percutaneous Approach-eluting | |
| Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Radial Artery with Two Drug-eluting | |
| Intraluminal Devices, Percutaneous Approach-eluting | |
| Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Radial Artery, Bifurcation, with Three Drug- | |
| eluting Intraluminal Devices, Percutaneous Approach-eluting | |
| Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Radial Artery with Three Drug-eluting | |
| Dilation of Left Radial Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting | |
| | eluting Intraluminal Devices, Open Approach-eluting Intraluminal Devices, Open Approach Dilation of Left Radial Artery, Bifurcation, with Intraluminal Device, Open Approach— Dilation of Left Radial Artery with Intraluminal Device, Open Approach— Dilation of Left Radial Artery, Bifurcation, with Two Intraluminal Devices, Open Approach— Dilation of Left Radial Artery with Two Intraluminal Devices, Open Approach— Dilation of Left Radial Artery, Bifurcation, with Three Intraluminal Devices, Open Approach— Dilation of Left Radial Artery with Three Intraluminal Devices, Open Approach— Dilation of Left Radial Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach— Dilation of Left Radial Artery with Four or More Intraluminal Devices, Open Approach— Dilation of Left Radial Artery, Bifurcation, Open Approach— Dilation of Left Radial Artery, Bifurcation, Open Approach— Dilation of Left Radial Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Radial Artery with Drug-eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Radial Artery with Drug-eluting Intraluminal Device, Percutaneous Approach Dilation of Left Radial Artery, Bifurcation, with Two Drug- eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Radial Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Radial Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting |


| | Poulsion of Extraluminal Device in Lower Vein Deventer | |
|---|---|---|
| 06\4\7467 | Revision of Extraluminal Device in Lower Vein, Percutaneous | |
| 06WY4CZ | Endoscopic Approach— Revision of Intraluminal Device in Lower Vein, Percutaneous | |
| 06WY4DZ | Endoscopic Approach— | |
| HCPCS | | |
| 35256 | | |
| 35286 | | |
| 35351 | | |
| 35355 | | |
| 35361 | | |
| 35363 | | |
| 35371 | | |
| 35372 | | |
| 35381 | | |
| 35454 | | |
| 35456 | | |
| 35459 | | |
| 35470 | | |
| 35473 | | |
| 35474 | | |
| 35482 | | |
| 35483 | | |
| 35485 | | |
| 35492 | | |
| 35493 | | |
| 35495 | | |
| 35521 | | |
| 35533 | | |
| 35556 | | |
| 35558 | | |
| 35563 | | |
| 35565 | | |
| 35566 | | |
| 35571 | | |
| 35621 | | |
| 35623 | | |
| 35641 | | |
| 35646 | | |
| 35647 | | |
| 35650 | | |
| 35651 | | |
| 35654 | | |
| 35656 | | |
| 35661 | | |
| 35663 | | |
| 35666 | | |
| 35671 | | |
| Hypertension | | |
| ICD10 Dx | CD9 Dx LongDesiCD10 Long | pDesICD9 |
| · | | · |

582

| 110 | 1010 | le | las is a second of the second |
|---|---|---|---|
| 110 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| <u> </u> | 4011<br>4019 | Essential (primary) hypertension | Benign essential hypertension Unspecified essential hypertension |
| 1160 | 4019 | Essential (primary) hypertension Hypertensive urgency | Unspecified essential hypertension |
| 1161 | 4019 | Hypertensive digency Hypertensive emergency | Unspecified essential hypertension |
| 1169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| 1119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| l110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| 1110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| l110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage I through stage IV, or unspecified |
| I120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| 1129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage I |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| .255 | .0.01 | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| 11311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| 11311 | 10 102 | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| 1132 | 40403 | , · · | with heart failure and with chronic kidney disease stage V or |
| | | failure and with stage 5 chronic kidney disease, or end stage | |
| 11210 | 40410 | renal disease | end stage renal disease |
| 11310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage I |
| 1422 | 40444 | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I through |
| | | or unspecified chronic kidney disease | stage IV, or unspecified |
| 11311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| I132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end stage | heart failure and chronic kidney disease stage V or end stage |
| | | renal disease | renal disease |
| 11310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage I |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| L | | . ~ | . · |

| l132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
|---|---|---|---|
| | | failure and with stage 5 chronic kidney disease, or end stage | with heart failure and chronic kidney disease stage V or end |
| | | renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| I150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| I151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| I152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| I158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| I159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

Diabetes


Hyperlipidem ia

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| E780 | 2720 | Pure hypercholesterolemia | PURE HYPERCHOLESTEROLEMIA |
| E7800 | 2722 | | MIXED HYPERLIPIDEMIA |
| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| M10372 | 40410 | Gout due to renal impairment, left ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
|---|---|---|---|
| | | | BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M10379 | 40411 | Gout due to renal impairment, unspecified ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M1038 | 40412 | Gout due to renal impairment, vertebrae | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M1039 | 40413 | Gout due to renal impairment, multiple sites | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M3214 | 4049 | Glomerular disease in systemic lupus erythematosus | UNSPECIFIED HYPERTENSIVE HEART AND KIDNEY DISEASE |
| M3215 | 40490 | Tubulo-interstitial nephropathy in systemic lupus | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | erythematosus | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | · · | KIDNEY DISEASE STAGE I THROUGH STAGE IV OR |
| | | | UNSPECIFIED |
| M3504 | 40491 | Sicca syndrome with tubulo-interstitial nephropathy | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| 1413304 | 40431 | Sieca syndrome with tubulo interstitial hepinopathy | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| NOOO | 40402 | A - 1 | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| N000 | 40492 | Acute nephritic syndrome with minor glomerular | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | abnormality | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | | KIDNEY DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N001 | 40493 | Acute nephritic syndrome with focal and segmental | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | glomerular lesions | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N002 | 4533 | Acute nephritic syndrome with diffuse membranous | EMBOLISM AND THROMBOSIS OF RENAL VEIN |
| | | glomerulonephritis | |
| N003 | 5800 | Acute nephritic syndrome with diffuse mesangial | ACUTE GLOMERULONEPHRITIS WITH LESION OF |
| | | proliferative glomerulonephritis | PROLIFERATIVE GLOMERULONEPHRITIS |
| N004 | 5804 | Acute nephritic syndrome with diffuse endocapillary | ACUTE GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | proliferative glomerulonephritis | PROGRESSIVE GLOMERULONEPHRITIS |
| N005 | 5808 | Acute nephritic syndrome with diffuse mesangiocapillary | ACUTE GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| .1005 | 5000 | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N006 | 5809 | Acute nephritic syndrome with dense deposit disease | ACUTE GLOMERULONEPHRITIS WITH UNSPECIFIED |
| 14000 | 3003 | Acute hepilitie syndrome with dense deposit disease | PATHOLOGICAL LESION IN KIDNEY |
| N007 | 581 | Acute nephritic syndrome with diffuse crescentic | NEPHROTIC SYNDROME |
| 11007 | 301 | glomerulonephritis | NEPHROTIC STNDROWIE |
| NOOO | 5040 | | NEDUDOTIC CVAIDDOMAE MUTULESCOM OF BROUFERATIVE |
| N008 | 5810 | Acute nephritic syndrome with other morphologic changes | NEPHROTIC SYNDROME WITH LESION OF PROLIFERATIVE |
| ***** | 5044 | | GLOMERULONEPHRITIS |
| N009 | 5811 | Acute nephritic syndrome with unspecified morphologic | NEPHROTIC SYNDROME WITH LESION OF MEMBRANOUS |
| | | changes | GLOMERULONEPHRITIS |
| N010 | 5812 | Rapidly progressive nephritic syndrome with minor | NEPHROTIC SYNDROME WITH LESION OF |
| | | glomerular abnormality | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N011 | 5813 | Rapidly progressive nephritic syndrome with focal and | NEPHROTIC SYNDROME WITH LESION OF MINIMAL CHANG |
| | | segmental glomerular lesions | GLOMERULONEPHRITIS |
| N012 | 5818 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH OTHER SPECIFIED |
| | | membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N013 | 58181 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME IN DISEASES CLASSIFIED |
| | | mesangial proliferative glomerulonephritis | ELSEWHERE |
| N014 | 58189 | Rapidly progressive nephritic syndrome with diffuse | OTHER NEPHROTIC SYNDROME WITH SPECIFIED |
| - '- | | endocapillary proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED PATHOLOGICAL |
| | 3023 | mesangiocapillary glomerulonephritis | LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense deposit | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| INOTO | 3020 | | |
| NC47 | 5021 | disease | PROLIFERATIVE GLOMERULONEPHRITIS |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | CHRONIC GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| 11013 | | | |

| N020 | 5828 | Recurrent and persistent hematuria with minor glomerular | CHRONIC GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
|---|---|---|---|
| | | abnormality | PATHOLOGICAL LESION IN KIDNEY |
| N021 | 5829 | Recurrent and persistent hematuria with focal and | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED |
| | | segmental glomerular lesions | PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | membranous glomerulonephritis | OR CHRONIC WITH LESION OF PROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N023 | 5831 | Recurrent and persistent hematuria with diffuse mesangial | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOUS |
| | | | GLOMERULONEPHRITIS |
| N024 | 5832 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | endocapillary proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOPROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | mesangiocapillary glomerulonephritis | OR CHRONIC WITH LESION OF RAPIDLY PROGRESSIVE |
| | | | GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | disease | OR CHRONIC WITH LESION OF RENAL CORTICAL NECROSIS |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse crescentic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | glomerulonephritis | OR CHRONIC WITH LESION OF RENAL MEDULLARY NECROS |
| N028 | 5838 | Recurrent and persistent hematuria with other morphologic | |
| | | changes | OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESION |
| | | | IN KIDNEY |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | morphologic changes | OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN |
| | | | KIDNEY |
| N030 | 5846 | Chronic nephritic syndrome with minor glomerular | ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICA |
| | | abnormality | NECROSIS |
| N031 | 5847 | Chronic nephritic syndrome with focal and segmental | ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLA |
| | | glomerular lesions | (PAPILLARY) NECROSIS |
| N032 | 5848 | Chronic nephritic syndrome with diffuse membranous | ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED |
| | | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N033 | 5849 | Chronic nephritic syndrome with diffuse mesangial | ACUTE KIDNEY FAILURE UNSPECIFIED |
| | | proliferative glomerulonephritis | |
| N034 | 5851 | Chronic nephritic syndrome with diffuse endocapillary | CHRONIC KIDNEY DISEASE STAGE I |
| | | proliferative glomerulonephritis | |
| N035 | 5852 | Chronic nephritic syndrome with diffuse mesangiocapillary | CHRONIC KIDNEY DISEASE STAGE II (MILD) |
| | | glomerulonephritis | |
| N036 | 5853 | Chronic nephritic syndrome with dense deposit disease | CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N037 | 5854 | Chronic nephritic syndrome with diffuse crescentic | CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| | | glomerulonephritis | |
| N038 | 5855 | Chronic nephritic syndrome with other morphologic changes | CHRONIC KIDNEY DISEASE STAGE V |
| N039 | 5856 | Chronic nephritic syndrome with unspecified morphologic | END STAGE RENAL DISEASE |
| | | changes | |
| N040 | 5859 | Nephrotic syndrome with minor glomerular abnormality | CHRONIC KIDNEY DISEASE UNSPECIFIED |
| N041 | 86600 | Nephrotic syndrome with focal and segmental glomerular | UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND |
| | | lesions | INTO CAVITY |
| N042 | 86601 | Nephrotic syndrome with diffuse membranous | HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE |
| | | glomerulonephritis | WITHOUT OPEN WOUND INTO CAVITY |
| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative | INJURY TO KIDNEY WITH OPEN WOUND INTO CAVITY |
| | | glomerulonephritis | |
| N044 | | Nephrotic syndrome with diffuse endocapillary proliferative | |
| | | glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic | |
| | | glomerulonephritis | |
| N048 | | Nephrotic syndrome with other morphologic changes | |
| N049 | I | Nephrotic syndrome with unspecified morphologic changes | |

| | | T |
|---|---|---|
| N050 | Unspecified nephritic syndrome with minor glomerular | |
| NOE1 | abnormality | |
| N051 | Unspecified nephritic syndrome with focal and segmental glomerular lesions | |
| N052 | Unspecified nephritic syndrome with diffuse membranous | |
| | glomerulonephritis | |
| N053 | Unspecified nephritic syndrome with diffuse mesangial | |
| | proliferative glomerulonephritis | |
| N054 | Unspecified nephritic syndrome with diffuse endocapillary | |
| 11054 | proliferative glomerulonephritis | |
| N055 | Unspecified nephritic syndrome with diffuse | |
| 14055 | mesangiocapillary glomerulonephritis | |
| N056 | Unspecified nephritic syndrome with dense deposit disease | |
| N057 | Unspecified nephritic syndrome with diffuse crescentic | |
| INU57 | | |
| NOTO | glomerulonephritis | |
| N058 | Unspecified nephritic syndrome with other morphologic | |
| | changes | |
| N059 | Unspecified nephritic syndrome with unspecified | |
| | morphologic changes | |
| N060 | Isolated proteinuria with minor glomerular abnormality | |
| N061 | Isolated proteinuria with focal and segmental glomerular | |
| | lesions | |
| N062 | Isolated proteinuria with diffuse membranous | |
| | glomerulonephritis | |
| N063 | Isolated proteinuria with diffuse mesangial proliferative | |
| | glomerulonephritis | |
| N064 | Isolated proteinuria with diffuse endocapillary proliferative | |
| | glomerulonephritis | |
| N065 | Isolated proteinuria with diffuse mesangiocapillary | |
| | glomerulonephritis | |
| N066 | Isolated proteinuria with dense deposit disease | |
| N067 | Isolated proteinuria with diffuse crescentic | |
| | glomerulonephritis | |
| N068 | Isolated proteinuria with other morphologic lesion | |
| N069 | Isolated proteinuria with unspecified morphologic lesion | |
| N070 | Hereditary nephropathy, not elsewhere classified with | |
| | minor glomerular abnormality | |
| N071 | Hereditary nephropathy, not elsewhere classified with focal | |
| | and segmental glomerular lesions | |
| N072 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse membranous glomerulonephritis | |
| N073 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangial proliferative glomerulonephritis | |
| N074 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse endocapillary proliferative glomerulonephritis | |
| N075 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangiocapillary glomerulonephritis | |
| N076 | Hereditary nephropathy, not elsewhere classified with | |
| 1,0,0 | dense deposit disease | |
| N077 | Hereditary nephropathy, not elsewhere classified with | |
| , | diffuse crescentic glomerulonephritis | |
| N078 | Hereditary nephropathy, not elsewhere classified with | |
| 1,070 | other morphologic lesions | |
| N079 | Hereditary nephropathy, not elsewhere classified with | |
| 14075 | unspecified morphologic lesions | |
| N08 | Glomerular disorders in diseases classified elsewhere | |
| N140 | Analgesic nephropathy Nephropathy indused by other drugs medicaments and | |
| N141 | Nephropathy induced by other drugs, medicaments and | |
| N14.63 | biological substances | |
| N142 | Nephropathy induced by unspecified drug, medicament or | |
| N14.63 | biological substance | |
| N143 | Nephropathy induced by heavy metals | |


## Appendix A Comorbid conditions

| 90964 |
|-------|
| 90965 |
| 90966 |
| 90967 |
| 90968 |
| 90969 |
| 90970 |
| 90989 |
| 90993 |
| 99512 |
| 99559 |

Chronic liver disease


## Appendix A Comorbid conditions

| K7581 | Nonalcoholic steatohepatitis (NASH) |
|-------|---------------------------------------------------|
| K7589 | Other specified inflammatory liver diseases |
| K759 | Inflammatory liver disease, unspecified |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K761 | Chronic passive congestion of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K765 | Hepatic veno-occlusive disease |
| K766 | Portal hypertension |
| K767 | Hepatorenal syndrome |
| K7681 | Hepatopulmonary syndrome |
| K7689 | Other specified diseases of liver |
| K769 | Liver disease, unspecified |
| K77 | Liver disorders in diseases classified elsewhere |

## **Asthma**


Ischemic heart disease


## Appendix A Comorbid conditions


COPD

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| J40 | 490 | Bronchitis, not specified as acute or chronic | BRONCHITIS NOT SPECIFIED AS ACUTE OR CHRONIC |
| J410 | 491 | Simple chronic bronchitis | CHRONIC BRONCHITIS |
| J411 | 4910 | Mucopurulent chronic bronchitis | SIMPLE CHRONIC BRONCHITIS |
| J418 | 4911 | Mixed simple and mucopurulent chronic bronchitis | MUCOPURULENT CHRONIC BRONCHITIS |
| J42 | 4912 | Unspecified chronic bronchitis | OBSTRUCTIVE CHRONIC BRONCHITIS |
| J430 | 49120 | Unilateral pulmonary emphysema [MacLeod's syndrome] | OBSTRUCTIVE CHRONIC BRONCHITIS WITHOUT |
| | | | EXACERBATION |
| J431 | 49121 | Panlobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH (ACUTE) |
| | | | EXACERBATION |
| J432 | 49122 | Centrilobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH ACUTE |
| | | | BRONCHITIS |
| J438 | 4918 | Other emphysema | OTHER CHRONIC BRONCHITIS |
| J439 | 4919 | Emphysema, unspecified | UNSPECIFIED CHRONIC BRONCHITIS |
| J440 | 492 | Chronic obstructive pulmonary disease with acute lower | EMPHYSEMA |
| | | respiratory infection | |
| J441 | 4920 | Chronic obstructive pulmonary disease with (acute) | EMPHYSEMATOUS BLEB |
| | | exacerbation | |
| J449 | 4928 | Chronic obstructive pulmonary disease, unspecified | OTHER EMPHYSEMA |
| J470 | 494 | Bronchiectasis with acute lower respiratory infection | BRONCHIECTASIS |
| J471 | 4940 | Bronchiectasis with (acute) exacerbation | BRONCHIECTASIS WITHOUT ACUTE EXACERBATION |
| J479 | 4941 | Bronchiectasis, uncomplicated | BRONCHIECTASIS WITH ACUTE EXACERBATION |
| | 496 | | CHRONIC AIRWAY OBSTRUCTION NOT ELSEWHERE |
| | | | CLASSIFIED |

Occurence of malignancy

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| C000 | 140 | Malignant neoplasm of external upper lip | MALIGNANT NEOPLASM OF LIP |
| C001 | 1400 | Malignant neoplasm of external lower lip | MALIGNANT NEOPLASM OF UPPER LIP VERMILION BORDER |
| C002 | 1401 | Malignant neoplasm of external lip, unspecified | MALIGNANT NEOPLASM OF LOWER LIP VERMILION BORDER |
| C003 | 1403 | Malignant neoplasm of upper lip, inner aspect | MALIGNANT NEOPLASM OF UPPER LIP INNER ASPECT |
| C004 | 1404 | Malignant neoplasm of lower lip, inner aspect | MALIGNANT NEOPLASM OF LOWER LIP INNER ASPECT |
| C005 | 1405 | Malignant neoplasm of lip, unspecified, inner aspect | MALIGNANT NEOPLASM OF LIP UNSPECIFIED INNER ASPECT |
| C006 | 1406 | Malignant neoplasm of commissure of lip, unspecified | MALIGNANT NEOPLASM OF COMMISSURE OF LIP |
| C008 | 1408 | Malignant neoplasm of overlapping sites of lip | MALIGNANT NEOPLASM OF OTHER SITES OF LIP |
| C009 | 1409 | Malignant neoplasm of lip, unspecified | MALIGNANT NEOPLASM OF LIP UNSPECIFIED VERMILION |
| | | | BORDER |
| C01 | 141 | Malignant neoplasm of base of tongue | MALIGNANT NEOPLASM OF TONGUE |
| C020 | 1410 | Malignant neoplasm of dorsal surface of tongue | MALIGNANT NEOPLASM OF BASE OF TONGUE |
| C021 | 1411 | Malignant neoplasm of border of tongue | MALIGNANT NEOPLASM OF DORSAL SURFACE OF TONGUE |
| C022 | 1412 | Malignant neoplasm of ventral surface of tongue | MALIGNANT NEOPLASM OF TIP AND LATERAL BORDER OF |
| | | | TONGUE |

| C023 | 1413 | Malignant neoplasm of anterior two-thirds of tongue, part unspecified | MALIGNANT NEOPLASM OF VENTRAL SURFACE OF TONGUE |
|---|---|---|---|
| C024 | 1414 | Malignant neoplasm of lingual tonsil | MALIGNANT NEOPLASM OF ANTERIOR TWO-THIRDS OF TONGUE PART UNSPECIFIED |
| C028 | 1415 | Malignant neoplasm of overlapping sites of tongue | MALIGNANT NEOPLASM OF JUNCTIONAL ZONE OF TONGUE |
| C029 | 1416 | Malignant neoplasm of tongue, unspecified | MALIGNANT NEOPLASM OF LINGUAL TONSIL |
| C030 | 1418 | Malignant neoplasm of upper gum | MALIGNANT NEOPLASM OF OTHER SITES OF TONGUE |
| C031 | 1419 | Malignant neoplasm of lower gum | MALIGNANT NEOPLASM OF TONGUE UNSPECIFIED |
| C039 | 142 | Malignant neoplasm of gum, unspecified | MALIGNANT NEOPLASM OF MAJOR SALIVARY GLANDS |
| C040 | 1420 | Malignant neoplasm of anterior floor of mouth | MALIGNANT NEOPLASM OF PAROTID GLAND |
| C041 | 1421 | Malignant neoplasm of lateral floor of mouth | MALIGNANT NEOPLASM OF SUBMANDIBULAR GLAND |
| C048 | 1422 | Malignant neoplasm of overlapping sites of floor of mouth | MALIGNANT NEOPLASM OF SUBLINGUAL GLAND |
| C049 | 1428 | Malignant neoplasm of floor of mouth, unspecified | MALIGNANT NEOPLASM OF OTHER MAJOR SALIVARY GLANDS |
| C050 | 1429 | Malignant neoplasm of hard palate | MALIGNANT NEOPLASM OF SALIVARY GLAND UNSPECIFIED |
| C051 | 143 | Malignant neoplasm of soft palate | MALIGNANT NEOPLASM OF GUM |
| C052 | 1430 | Malignant neoplasm of uvula | MALIGNANT NEOPLASM OF UPPER GUM |
| C058 | 1431 | Malignant neoplasm of overlapping sites of palate | MALIGNANT NEOPLASM OF LOWER GUM |
| C059 | 1438 | Malignant neoplasm of palate, unspecified | MALIGNANT NEOPLASM OF OTHER SITES OF GUM |
| C060 | 1439 | Malignant neoplasm of cheek mucosa | MALIGNANT NEOPLASM OF GUM UNSPECIFIED |
| C061 | 144 | Malignant neoplasm of vestibule of mouth | MALIGNANT NEOPLASM OF FLOOR OF MOUTH |
| C062 | 1440 | Malignant neoplasm of retromolar area | MALIGNANT NEOPLASM OF ANTERIOR PORTION OF FLOOR OF MOUTH |
| C0680 | 1441 | Malignant neoplasm of overlapping sites of unspecified parts of mouth | MALIGNANT NEOPLASM OF LATERAL PORTION OF FLOOR OF MOUTH |
| C0689 | 1448 | Malignant neoplasm of overlapping sites of other parts of mouth | MALIGNANT NEOPLASM OF OTHER SITES OF FLOOR OF MOUTH |
| C069 | 1449 | Malignant neoplasm of mouth, unspecified | MALIGNANT NEOPLASM OF FLOOR OF MOUTH PART UNSPECIFIED |
| C07 | 145 | Malignant neoplasm of parotid gland | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF MOUTH |
| C080 | 1450 | Malignant neoplasm of submandibular gland | MALIGNANT NEOPLASM OF CHEEK MUCOSA |
| C081 | 1451 | Malignant neoplasm of sublingual gland | MALIGNANT NEOPLASM OF VESTIBULE OF MOUTH |
| C089 | 1452 | Malignant neoplasm of major salivary gland, unspecified | MALIGNANT NEOPLASM OF HARD PALATE |
| C090 | 1453 | Malignant neoplasm of tonsillar fossa | MALIGNANT NEOPLASM OF SOFT PALATE |
| C091 | 1454 | Malignant neoplasm of tonsillar pillar (anterior) (posterior) | MALIGNANT NEOPLASM OF UVULA |
| C098 | 1455 | Malignant neoplasm of overlapping sites of tonsil | MALIGNANT NEOPLASM OF PALATE UNSPECIFIED |
| C099 | 1456 | Malignant neoplasm of tonsil, unspecified | MALIGNANT NEOPLASM OF RETROMOLAR AREA |
| C100 | 1458 | Malignant neoplasm of vallecula | MALIGNANT NEOPLASM OF OTHER SPECIFIED PARTS OF MOUTH |
| C101 | 1459 | Malignant neoplasm of anterior surface of epiglottis | MALIGNANT NEOPLASM OF MOUTH UNSPECIFIED |
| C102 | 146 | Malignant neoplasm of lateral wall of oropharynx | MALIGNANT NEOPLASM OF OROPHARYNX |
| C103 | 1460 | Malignant neoplasm of posterior wall of oropharynx | MALIGNANT NEOPLASM OF TONSIL |
| C104 | 1461 | Malignant neoplasm of branchial cleft | MALIGNANT NEOPLASM OF TONSILLAR FOSSA |
| C108 | 1462 | Malignant neoplasm of overlapping sites of oropharynx | MALIGNANT NEOPLASM OF TONSILLAR PILLARS (ANTERIOR) (POSTERIOR) |
| C109 | 1463 | Malignant neoplasm of oropharynx, unspecified | MALIGNANT NEOPLASM OF VALLECULA EPIGLOTTICA |
| C110 | 1464 | Malignant neoplasm of superior wall of nasopharynx | MALIGNANT NEOPLASM OF ANTERIOR ASPECT OF EPIGLOTTIS |
| C111 | 1465 | Malignant neoplasm of posterior wall of nasopharynx | MALIGNANT NEOPLASM OF JUNCTIONAL REGION OF OROPHARYNX |
| C112 | 1466 | Malignant neoplasm of lateral wall of nasopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF<br>OROPHARYNX |
| C113 | 1467 | Malignant neoplasm of anterior wall of nasopharynx | MALIGNANT NEOPLASM OF POSTERIOR WALL OF OROPHARYNX |
| C118 | 1468 | Malignant neoplasm of overlapping sites of nasopharynx | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF OROPHARYNX |
| C119 | 1469 | Malignant neoplasm of nasopharynx, unspecified | MALIGNANT NEOPLASM OF OROPHARYNX UNSPECIFIED SITE |
| C12 | 147 | Malignant neoplasm of pyriform sinus | MALIGNANT NEOPLASM OF NASOPHARYNX |
| C130 | 1470 | Malignant neoplasm of postcricoid region | MALIGNANT NEOPLASM OF SUPERIOR WALL OF |
|---|---|---|---|
| | | | NASOPHARYNX |
| C131 | 1471 | Malignant neoplasm of aryepiglottic fold, hypopharyngeal aspect | MALIGNANT NEOPLASM OF POSTERIOR WALL OF NASOPHARYNX |
| C132 | 1472 | Malignant neoplasm of posterior wall of hypopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF NASOPHARYNX |
| C138 | 1473 | Malignant neoplasm of overlapping sites of hypopharynx | MALIGNANT NEOPLASM OF ANTERIOR WALL OF |
| C130 | 1175 | Wanghane neoplasm of overlapping siees of mypopharym | NASOPHARYNX |
| C139 | 1478 | Malignant neoplasm of hypopharynx, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | , , , , , , | NASOPHARYNX |
| C140 | 1479 | Malignant neoplasm of pharynx, unspecified | MALIGNANT NEOPLASM OF NASOPHARYNX UNSPECIFIED SITE |
| C142 | 148 | Malignant neoplasm of Waldeyer's ring | MALIGNANT NEOPLASM OF HYPOPHARYNX |
| C148 | 1480 | Malignant neoplasm of overlapping sites of lip, oral cavity | MALIGNANT NEOPLASM OF POSTCRICOID REGION OF |
| | | and pharynx | HYPOPHARYNX |
| C153 | 1481 | Malignant neoplasm of upper third of esophagus | MALIGNANT NEOPLASM OF PYRIFORM SINUS |
| C154 | 1482 | Malignant neoplasm of middle third of esophagus | MALIGNANT NEOPLASM OF ARYEPIGLOTTIC FOLD |
| | | | HYPOPHARYNGEAL ASPECT |
| C155 | 1483 | Malignant neoplasm of lower third of esophagus | MALIGNANT NEOPLASM OF POSTERIOR HYPOPHARYNGEAL |
| | | | WALL |
| C158 | 1488 | Malignant neoplasm of overlapping sites of esophagus | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | HYPOPHARYNX |
| C159 | 1489 | Malignant neoplasm of esophagus, unspecified | MALIGNANT NEOPLASM OF HYPOPHARYNX UNSPECIFIED |
| | | | SITE |
| C160 | 149 | Malignant neoplasm of cardia | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES |
| | | | WITHIN THE LIP ORAL CAVITY AND PHARYNX |
| C161 | 1490 | Malignant neoplasm of fundus of stomach | MALIGNANT NEOPLASM OF PHARYNX UNSPECIFIED |
| C162 | 1491 | Malignant neoplasm of body of stomach | MALIGNANT NEOPLASM OF WALDEYER'S RING |
| C163 | 1498 | Malignant neoplasm of pyloric antrum | MALIGNANT NEOPLASM OF OTHER SITES WITHIN THE LIP |
| | | | AND ORAL CAVITY |
| C164 | 1499 | Malignant neoplasm of pylorus | MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE |
| | | | LIP AND ORAL CAVITY |
| C165 | 150 | Malignant neoplasm of lesser curvature of stomach, unspecified | MALIGNANT NEOPLASM OF ESOPHAGUS |
| C166 | 1500 | Malignant neoplasm of greater curvature of stomach, unspecified | MALIGNANT NEOPLASM OF CERVICAL ESOPHAGUS |
| C168 | 1501 | Malignant neoplasm of overlapping sites of stomach | MALIGNANT NEOPLASM OF THORACIC ESOPHAGUS |
| C169 | 1502 | Malignant neoplasm of stomach, unspecified | MALIGNANT NEOPLASM OF ABDOMINAL ESOPHAGUS |
| C170 | 1503 | Malignant neoplasm of duodenum | MALIGNANT NEOPLASM OF UPPER THIRD OF ESOPHAGUS |
| C171 | 1504 | Malignant neoplasm of jejunum | MALIGNANT NEOPLASM OF MIDDLE THIRD OF ESOPHAGUS |
| C172 | 1505 | Malignant neoplasm of ileum | MALIGNANT NEOPLASM OF LOWER THIRD OF ESOPHAGUS |
| C173 | 1508 | Meckel's diverticulum, malignant | MALIGNANT NEOPLASM OF OTHER SPECIFIED PART OF |
| | | The state of the s | ESOPHAGUS |
| C178 | 1509 | Malignant neoplasm of overlapping sites of small intestine | MALIGNANT NEOPLASM OF ESOPHAGUS UNSPECIFIED SITE |
| C179 | 151 | Malignant neoplasm of small intestine, unspecified | MALIGNANT NEOPLASM OF STOMACH |
| C180 | 1510 | Malignant neoplasm of cecum | MALIGNANT NEOPLASM OF CARDIA |
| C181 | 1511 | Malignant neoplasm of appendix | MALIGNANT NEOPLASM OF PYLORUS |
| C182 | 1512 | Malignant neoplasm of ascending colon | MALIGNANT NEOPLASM OF PYLORIC ANTRUM |
| C183 | 1513 | Malignant neoplasm of hepatic flexure | MALIGNANT NEOPLASM OF FUNDUS OF STOMACH |
| C184 | 1514 | Malignant neoplasm of transverse colon | MALIGNANT NEOPLASM OF BODY OF STOMACH |
| C185 | 1515 | Malignant neoplasm of splenic flexure | MALIGNANT NEOPLASM OF LESSER CURVATURE OF |
| | | | STOMACH UNSPECIFIED |
| C186 | 1516 | Malignant neoplasm of descending colon | MALIGNANT NEOPLASM OF GREATER CURVATURE OF |
| | | J | STOMACH UNSPECIFIED |
| C187 | 1518 | Malignant neoplasm of sigmoid colon | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| - | | | STOMACH |
| C188 | 1519 | Malignant neoplasm of overlapping sites of colon | MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED SITE |
| C189 | 152 | Malignant neoplasm of colon, unspecified | MALIGNANT NEOPLASM OF SMALL INTESTINE INCLUDING |
| | | | DUODENUM |
| C19 | 1520 | Malignant neoplasm of rectosigmoid junction | MALIGNANT NEOPLASM OF DUODENUM |

| C20 | 1521 | Malignant neoplasm of rectum | MALIGNANT NEOPLASM OF JEJUNUM |
|---|---|---|---|
| C210 | 1522 | Malignant neoplasm of anus, unspecified | MALIGNANT NEOPLASM OF ILEUM |
| C211 | 1523 | Malignant neoplasm of anal canal | MALIGNANT NEOPLASM OF MECKEL'S DIVERTICULUM |
| C212 | 1528 | Malignant neoplasm of cloacogenic zone | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| CLIL | 1320 | Manghane neophasm of diodeogetine zone | SMALL INTESTINE |
| C218 | 1529 | Malignant neoplasm of overlapping sites of rectum, anus | MALIGNANT NEOPLASM OF SMALL INTESTINE UNSPECIFIED |
| CLIC | 1323 | and anal canal | ISITE |
| C220 | 153 | Liver cell carcinoma | MALIGNANT NEOPLASM OF COLON |
| C221 | 1530 | Intrahepatic bile duct carcinoma | MALIGNANT NEOPLASM OF HEPATIC FLEXURE |
| C222 | 1531 | Hepatoblastoma | MALIGNANT NEOPLASM OF TRANSVERSE COLON |
| C223 | 1532 | Angiosarcoma of liver | MALIGNANT NEOPLASM OF DESCENDING COLON |
| C224 | 1533 | Other sarcomas of liver | MALIGNANT NEOPLASM OF SIGMOID COLON |
| C227 | 1534 | Other specified carcinomas of liver | MALIGNANT NEOPLASM OF CECUM |
| C228 | 1535 | Malignant neoplasm of liver, primary, unspecified as to type | |
| CZZO | 1555 | wanghant heopiasin of fiver, primary, anspeaned as to type | WALIGNAM NEOFEASW OF ATTEMOTO VERWIN ORIVIS |
| C229 | 1536 | Malignant neoplasm of liver, not specified as primary or | MALIGNANT NEOPLASM OF ASCENDING COLON |
| CZZJ | 1550 | secondary | WALIGNANT NEOF EASIN OF ASCENDING COLON |
| C23 | 1537 | Malignant neoplasm of gallbladder | MALIGNANT NEOPLASM OF SPLENIC FLEXURE |
| C240 | 1538 | Malignant neoplasm of extrahepatic bile duct | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C240 | 1556 | Walighant neoplasm of extranepatic bile duct | LARGE INTESTINE |
| C241 | 1539 | Malignant neoplasm of ampulla of Vater | MALIGNANT NEOPLASM OF COLON UNSPECIFIED SITE |
| C241<br>C248 | 1539 | Malignant neoplasm of overlapping sites of biliary tract | MALIGNANT NEOPLASM OF RECTUM RECTOSIGMOID |
| C246 | 154 | Manghant neoplasm of overlapping sites of billary tract | JUNCTION AND ANUS |
| C249 | 1540 | Malignant pooplasm of hillians tract, unspecified | MALIGNANT NEOPLASM OF RECTOSIGMOID JUNCTION |
| C249<br>C250 | 1540 | Malignant neoplasm of biliary tract, unspecified Malignant neoplasm of head of pancreas | MALIGNANT NEOPLASM OF RECTUM |
| | | Malignant neoplasm of body of pancreas | |
| C251 | 1542 | , , | MALIGNANT NEOPLASM OF ANAL CANAL |
| C252 | 1543 | Malignant neoplasm of tail of pancreas | MALIGNANT NEOPLASM OF ANUS UNSPECIFIED SITE |
| C253 | 1548 | Malignant neoplasm of pancreatic duct | MALIGNANT NEOPLASM OF OTHER SITES OF RECTUM |
| 625.4 | 455 | AA-P | RECTOSIGMOID JUNCTION AND ANUS |
| C254 | 155 | Malignant neoplasm of endocrine pancreas | MALIGNANT NEOPLASM OF LIVER AND INTRAHEPATIC BILE |
| 6257 | 4550 | Ad-Providence for the control of control | DUCTS |
| C257 | 1550 | Malignant neoplasm of other parts of pancreas | MALIGNANT NEOPLASM OF LIVER PRIMARY |
| C258 | 1551 | Malignant neoplasm of overlapping sites of pancreas | MALIGNANT NEOPLASM OF INTRAHEPATIC BILE DUCTS |
| C259 | 1552 | Malignant neoplasm of pancreas, unspecified | MALIGNANT NEOPLASM OF LIVER NOT SPECIFIED AS |
| 6260 | 456 | Malta and an afficial state of the state of | PRIMARY OR SECONDARY |
| C260 | 156 | Malignant neoplasm of intestinal tract, part unspecified | MALIGNANT NEOPLASM OF GALLBLADDER AND |
| 6264 | 4560 | AA-P | EXTRAHEPATIC BILE DUCTS |
| C261 | 1560 | Malignant neoplasm of spleen | MALIGNANT NEOPLASM OF GALLBLADDER |
| C269 | 1561 | Malignant neoplasm of ill-defined sites within the digestive | MALIGNANT NEOPLASM OF EXTRAHEPATIC BILE DUCTS |
| 6200 | 4562 | system | MANUCHANT NEODIACAA OF ANADIHLA OF WATER |
| C300 | 1562 | Malignant neoplasm of nasal cavity | MALIGNANT NEOPLASM OF AMPULLA OF VATER |
| C301 | 1568 | Malignant neoplasm of middle ear | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| 0240 | 4560 | AA II | GALLBLADDER AND EXTRAHEPATIC BILE DUCTS |
| C310 | 1569 | Malignant neoplasm of maxillary sinus | MALIGNANT NEOPLASM OF BILIARY TRACT PART |
| | | | UNSPECIFIED SITE |
| C311 | 157 | Malignant neoplasm of ethmoidal sinus | MALIGNANT NEOPLASM OF PANCREAS |
| C312 | 1570 | Malignant neoplasm of frontal sinus | MALIGNANT NEOPLASM OF HEAD OF PANCREAS |
| C313 | 1571 | Malignant neoplasm of sphenoid sinus | MALIGNANT NEOPLASM OF BODY OF PANCREAS |
| C318 | 1572 | Malignant neoplasm of overlapping sites of accessory | MALIGNANT NEOPLASM OF TAIL OF PANCREAS |
| | | sinuses | |
| C319 | 1573 | Malignant neoplasm of accessory sinus, unspecified | MALIGNANT NEOPLASM OF PANCREATIC DUCT |
| C320 | 1574 | Malignant neoplasm of glottis | MALIGNANT NEOPLASM OF ISLETS OF LANGERHANS |
| C321 | 1578 | Malignant neoplasm of supraglottis | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | PANCREAS |
| C322 | 1579 | Malignant neoplasm of subglottis | MALIGNANT NEOPLASM OF PANCREAS PART UNSPECIFIED |
| C323 | 158 | Malignant neoplasm of laryngeal cartilage | MALIGNANT NEOPLASM OF RETROPERITONEUM AND |
| | | | PERITONEUM |
| C328 | 1580 | Malignant neoplasm of overlapping sites of larynx | MALIGNANT NEOPLASM OF RETROPERITONEUM |
| C329 | 1588 | Malignant neoplasm of larynx, unspecified | MALIGNANT NEOPLASM OF SPECIFIED PARTS OF |
| | | | PERITONEUM |
| C33 | 1589 | Malignant neoplasm of trachea | MALIGNANT NEOPLASM OF PERITONEUM UNSPECIFIED |


| C438 | 1722 | Malignant melanoma of overlapping sites of skin | MALIGNANT MELANOMA OF SKIN OF EAR AND EXTERNAL |
|---|---|---|---|
| | | | AUDITORY CANAL |
| C439 | 1723 | Malignant melanoma of skin, unspecified | MALIGNANT MELANOMA OF SKIN OF OTHER AND UNSPECIFIED PARTS OF FACE |
| C450 | 1724 | Mesothelioma of pleura | MALIGNANT MELANOMA OF SKIN OF SCALP AND NECK |
| C451 | 1725 | Mesothelioma of peritoneum | MALIGNANT MELANOMA OF SKIN OF TRUNK EXCEPT SCROTUM |
| C452 | 1726 | Mesothelioma of pericardium | MALIGNANT MELANOMA OF SKIN OF UPPER LIMB INCLUDING SHOULDER |
| C457 | 1727 | Mesothelioma of other sites | MALIGNANT MELANOMA OF SKIN OF LOWER LIMB |
| C459 | 1728 | Mesothelioma, unspecified | MALIGNANT MELANOMA OF OTHER SPECIFIED SITES OF |
| C460 | 1729 | Kaposi's sarcoma of skin | SKIN |
| C460<br>C461 | 1729 | Kaposi's sarcoma of soft tissue | MELANOMA OF SKIN SITE UNSPECIFIED MALIGNANT NEOPLASM OF FEMALE BREAST |
| C461 | 1740 | | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF |
| | | Kaposi's sarcoma of palate | FEMALE BREAST |
| C463 | 1741 | Kaposi's sarcoma of lymph nodes | MALIGNANT NEOPLASM OF CENTRAL PORTION OF FEMALE BREAST |
| C464 | 1742 | Kaposi's sarcoma of gastrointestinal sites | MALIGNANT NEOPLASM OF UPPER-INNER QUADRANT OF FEMALE BREAST |
| C4650 | 1743 | Kaposi's sarcoma of unspecified lung | MALIGNANT NEOPLASM OF LOWER-INNER QUADRANT OF |
| | | | FEMALE BREAST |
| C4651 | 1744 | Kaposi's sarcoma of right lung | MALIGNANT NEOPLASM OF UPPER-OUTER QUADRANT OF |
| | | | FEMALE BREAST |
| C4652 | 1745 | Kaposi's sarcoma of left lung | MALIGNANT NEOPLASM OF LOWER-OUTER QUADRANT OF |
| | | | FEMALE BREAST |
| C467 | 1746 | Kaposi's sarcoma of other sites | MALIGNANT NEOPLASM OF AXILLARY TAIL OF FEMALE |
| C-107 | 1740 | Raposi s surcoma of other sites | BREAST |
| C469 | 1748 | Kaposi's sarcoma, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C 103 | 17 10 | haposi s surcoma, unspecimea | FEMALE BREAST |
| C470 | 1749 | Malignant neoplasm of peripheral nerves of head, face and | MALIGNANT NEOPLASM OF BREAST (FEMALE) UNSPECIFIED |
| C+70 | 1743 | neck | SITE |
| C4710 | 175 | Malignant neoplasm of peripheral nerves of unspecified | MALIGNANT NEOPLASM OF MALE BREAST |
| C4711 | 1750 | upper limb, including shoulder Malignant neoplasm of peripheral nerves of right upper | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF MALE |
| C4/11 | 1/50 | | BREAST |
| C4712 | 1750 | limb, including shoulder Malignant neoplasm of peripheral nerves of left upper limb, | |
| C4712 | 1759 | | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED SITE: |
| 04700 | 476 | including shoulder | OF MALE BREAST |
| C4720 | 176 | Malignant neoplasm of peripheral nerves of unspecified lower limb, including hip | KAPOSI'S SARCOMA |
| C4721 | 1760 | Malignant neoplasm of peripheral nerves of right lower limb, including hip | KAPOSI'S SARCOMA SKIN |
| C4722 | 1761 | Malignant neoplasm of peripheral nerves of left lower limb, including hip | KAPOSI'S SARCOMA SOFT TISSUE |
| | 1762 | | |
| C473 | 1/02 | Malignant neoplasm of peripheral nerves of thorax | KAPOSI'S SARCOMA PALATE |
| C474 | 1763 | Malignant neoplasm of peripheral nerves of abdomen | KAPOSI'S SARCOMA GASTROINTESTINAL SITES |
| | | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, | |
| C474<br>C475 | 1763<br>1764 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG |
| C474<br>C475<br>C476 | 1763<br>1764<br>1765 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES |
| C474<br>C475<br>C476<br>C478 | 1763<br>1764<br>1765<br>1768<br>1769 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE |
| C474<br>C475<br>C476<br>C478<br>C479 | 1763<br>1764<br>1765<br>1768<br>1769 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS |
| C474<br>C475<br>C476<br>C478<br>C479<br>C480<br>C481 | 1763<br>1764<br>1765<br>1768<br>1769<br>179<br>180 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum Malignant neoplasm of specified parts of peritoneum Malignant neoplasm of peritoneum, unspecified Malignant neoplasm of overlapping sites of retroperitoneum | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS MALIGNANT NEOPLASM OF CERVIX UTERI MALIGNANT NEOPLASM OF ENDOCERVIX |
| C474<br>C475<br>C476<br>C478<br>C479<br>C480<br>C481<br>C482 | 1763<br>1764<br>1765<br>1768<br>1769<br>179<br>180<br>1800 | Malignant neoplasm of peripheral nerves of abdomen Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, unspecified Malignant neoplasm of overlapping sites of peripheral nerves and autonomic nervous system Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified Malignant neoplasm of retroperitoneum Malignant neoplasm of specified parts of peritoneum Malignant neoplasm of peritoneum, unspecified | KAPOSI'S SARCOMA GASTROINTESTINAL SITES KAPOSI'S SARCOMA LUNG KAPOSI'S SARCOMA LYMPH NODES KAPOSI'S SARCOMA OTHER SPECIFIED SITES KAPOSI'S SARCOMA UNSPECIFIED SITE MALIGNANT NEOPLASM OF UTERUS-PART UNS MALIGNANT NEOPLASM OF CERVIX UTERI MALIGNANT NEOPLASM OF ENDOCERVIX |


| C50929 | 1909 | Malignant neoplasm of unspecified site of unspecified male breast | MALIGNANT NEOPLASM OF EYE PART UNSPECIFIED |
|---|---|---|---|
| C510 | 191 | Malignant neoplasm of labium majus | MALIGNANT NEOPLASM OF BRAIN |
| C511 | 1910 | Malignant neoplasm of labium minus | MALIGNANT NEOPLASM OF CEREBRUM EXCEPT LOBES AN VENTRICLES |
| C512 | 1911 | Malignant neoplasm of clitoris | MALIGNANT NEOPLASM OF FRONTAL LOBE |
| C518 | 1912 | Malignant neoplasm of overlapping sites of vulva | MALIGNANT NEOPLASM OF TEMPORAL LOBE |
| C519 | 1913 | Malignant neoplasm of vulva, unspecified | MALIGNANT NEOPLASM OF PARIETAL LOBE |
| C52 | 1914 | Malignant neoplasm of vagina | MALIGNANT NEOPLASM OF OCCIPITAL LOBE |
| C530 | 1915 | Malignant neoplasm of endocervix | MALIGNANT NEOPLASM OF VENTRICLES |
| C531 | 1916 | Malignant neoplasm of exocervix | MALIGNANT NEOPLASM OF CEREBELLUM NOT OTHERWIS |
| 0001 | 1510 | mang. and neephasm of electricity | SPECIFIED |
| C538 | 1917 | Malignant neoplasm of overlapping sites of cervix uteri | MALIGNANT NEOPLASM OF BRAIN STEM |
| C539 | 1918 | Malignant neoplasm of cervix uteri, unspecified | MALIGNANT NEOPLASM OF OTHER PARTS OF BRAIN |
| C540 | 1919 | Malignant neoplasm of isthmus uteri | MALIGNANT NEOPLASM OF BRAIN UNSPECIFIED SITE |
| C541 | 192 | Malignant neoplasm of endometrium | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF NERVOUS SYSTEM |
| C542 | 1920 | Malignant neoplasm of myometrium | MALIGNANT NEOPLASM OF CRANIAL NERVES |
| | | Malignant neoplasm of fundus uteri | MALIGNANT NEOPLASM OF CRANIAL NERVES MALIGNANT NEOPLASM OF CEREBRAL MENINGES |
| C543 | 1921 | · | |
| C548 | 1922 | Malignant neoplasm of overlapping sites of corpus uteri | MALIGNANT NEOPLASM OF SPINAL CORD |
| C549 | 1923 | Malignant neoplasm of corpus uteri, unspecified | MALIGNANT NEOPLASM OF SPINAL MENINGES |
| C55 | 1928 | Malignant neoplasm of uterus, part unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF NERVOUS SYSTEM |
| CEC1 | 1020 | Malignant needlasm of right overv | MALIGNANT NEOPLASM OF NERVOUS SYSTEM PART |
| C561 | 1929 | Malignant neoplasm of right ovary | UNSPECIFIED |
| CEGO | 102 | Malignant needless of left every | |
| C562 | 193 | Malignant neoplasm of left ovary | MALIGNANT NEOPLASM OF THYROID GLAND |
| C569 | 194 | Malignant neoplasm of unspecified ovary | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 05700 | 1010 | | AND RELATED STRUCTURES |
| C5700 | 1940 | Malignant neoplasm of unspecified fallopian tube | MALIGNANT NEOPLASM OF ADRENAL GLAND |
| C5701 | 1941 | Malignant neoplasm of right fallopian tube | MALIGNANT NEOPLASM OF PARATHYROID GLAND |
| C5702 | 1943 | Malignant neoplasm of left fallopian tube | MALIGNANT NEOPLASM OF PITUITARY GLAND AND |
| | | | CRANIOPHARYNGEAL DUCT |
| C5710 | 1944 | Malignant neoplasm of unspecified broad ligament | MALIGNANT NEOPLASM OF PINEAL GLAND |
| C5711 | 1945 | Malignant neoplasm of right broad ligament | MALIGNANT NEOPLASM OF CAROTID BODY |
| C5712 | 1946 | Malignant neoplasm of left broad ligament | MALIGNANT NEOPLASM OF AORTIC BODY AND OTHER PARAGANGLIA |
| C5720 | 1948 | Malignant neoplasm of unspecified round ligament | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 03720 | 25 .0 | manghant neophasin of anopeanica rouna ngament | AND RELATED STRUCTURES |
| C5721 | 1949 | Malignant neoplasm of right round ligament | MALIGNANT NEOPLASM OF ENDOCRINE GLAND SITE |
| C3721 | 1343 | Wanghane neoplasm of right Found ngament | UNSPECIFIED |
| C5722 | 195 | Malignant neoplasm of left round ligament | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITE |
| C573 | 1950 | Malignant neoplasm of parametrium | MALIGNANT NEOPLASM OF HEAD FACE AND NECK |
| C574 | 1951 | Malignant neoplasm of uterine adnexa, unspecified | MALIGNANT NEOPLASM OF THORAX |
| C577 | 1952 | Malignant neoplasm of other specified female genital organs | S MALIGNANT NEOPLASM OF ABDOMEN |
| C578 | 1953 | Malignant neoplasm of overlapping sites of female genital | MALIGNANT NEOPLASM OF PELVIS |
| C579 | 1954 | organs Malignant neoplasm of female genital organ, unspecified | MALIGNANT NEOPLASM OF UPPER LIMB |
| C579 | 1954 | Malignant neoplasm of lemale genital organ, unspecified Malignant neoplasm of placenta | MALIGNANT NEOPLASM OF LOWER LIMB |
| C600 | | Malignant neoplasm of prepuce | |
| | 1958 | Malignant neoplasm of prepuce Malignant neoplasm of glans penis | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| C601 | 196 | Mangnant neoplasm of glans penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM LYMPH NODES |
| C602 | 1960 | Malignant neoplasm of body of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 0000 | | | LYMPH NODES OF HEAD FACE AND NECK |
| C608 | 1961 | Malignant neoplasm of overlapping sites of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM INTRATHORACIC LYMPH NODES |
| C609 | 1962 | Malignant neoplasm of penis, unspecified | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 2233 | 1332 | | INTRA-ABDOMINAL LYMPH NODES |
| C61 | 1963 | Malignant neoplasm of prostate | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| COI | 1,000 | manghant neoplasm of prostate | SESSIONIL AND ONSI EGI IED MALIGINAMI MEOFEASIM |


| C7491 | 20071 | Malignant neoplasm of unspecified part of right adrenal | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF |
|---|---|---|---|
| | | gland | HEAD FACE AND NECK |
| C7492 | 20072 | Malignant neoplasm of unspecified part of left adrenal gland | LARGE CELL LYMPHOMA INVOLVING INTRATHORACIC LYMPH<br>NODES |
| C750 | 20073 | Malignant neoplasm of parathyroid gland | LARGE CELL LYMPHOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| C751 | 20074 | Malignant neoplasm of pituitary gland | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF |
| 6750 | 20075 | | AXILLA AND UPPER LIMB |
| C752 | 20075 | Malignant neoplasm of craniopharyngeal duct | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| C753 | 20076 | Malignant neoplasm of pineal gland | LARGE CELL LYMPHOMA INVOLVING INTRAPELVIC LYMPH NODES |
| C754 | 20077 | Malignant neoplasm of carotid body | LARGE CELL LYMPHOMA INVOLVING SPLEEN |
| C755 | 20078 | Malignant neoplasm of aortic body and other paraganglia | LARGE CELL LYMPHOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| C758 | 2008 | Malignant neoplasm with pluriglandular involvement, unspecified | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA |
| C759 | 20080 | Malignant neoplasm of endocrine gland, unspecified | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND |
| | | | RETICULOSARCOMA UNSPECIFIED SITE |
| C760 | 20081 | Malignant neoplasm of head, face and neck | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF HEAD FACE AND NECK |
| C761 | 20082 | Malignant neoplasm of thorax | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRATHORACIC LYMPH NODES |
| C762 | 20083 | Malignant neoplasm of abdomen | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRA-ABDOMINAL LYMPH NODES |
| C763 | 20084 | Malignant neoplasm of pelvis | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| C7640 | 20085 | Malignant neoplasm of unspecified upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF INGUINA REGION AND LOWER LIMB |
| C7641 | 20086 | Malignant neoplasm of right upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING INTRAPELVIC LYMPH NODES |
| C7642 | 20087 | Malignant neoplasm of left upper limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING SPLEEN |
| C7650 | 20088 | Malignant neoplasm of unspecified lower limb | OTHER NAMED VARIANTS OF LYMPHOSARCOMA AND RETICULOSARCOMA INVOLVING LYMPH NODES OF MULTIPLE SITES |
| C7651 | 201 | Malignant neoplasm of right lower limb | HODGKIN'S DISEASE |
| | 2010 | 0 1 0 | |
| C7652 | 1 | Malignant neoplasm of left lower limb | HODGKIN'S PARAGRANULOMA |
| C768<br>C770 | 20100<br>20101 | Malignant neoplasm of other specified ill-defined sites Secondary and unspecified malignant neoplasm of lymph | HODGKIN'S PARAGRANULOMA UNSPECIFIED SITE HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES |
| C771 | 20102 | nodes of head, face and neck Secondary and unspecified malignant neoplasm of | OF HEAD FACE AND NECK HODGKIN'S PARAGRANULOMA INVOLVING INTRATHORACIC |
| | | intrathoracic lymph nodes | LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING INTRA- |
| C772 | 20103 | Secondary and unspecified malignant neoplasm of intra- | HODOKIN STANAGIANOLOMA INVOLVING INTIA- |
| | | abdominal lymph nodes | ABDOMINAL LYMPH NODES |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES |
| C773 | 20104 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes Secondary and unspecified malignant neoplasm of | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB HODGKIN'S PARAGRANULOMA INVOLVING INTRAPELVIC |
| C773 C774 C775 | 20104<br>20105<br>20106 | abdominal lymph nodes Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes Secondary and unspecified malignant neoplasm of intrapelvic lymph nodes Secondary and unspecified malignant neoplasm of lymph | ABDOMINAL LYMPH NODES HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF AXILLA AND UPPER LIMB HODGKIN'S PARAGRANULOMA INVOLVING LYMPH NODES OF INGUINAL REGION AND LOWER LIMB HODGKIN'S PARAGRANULOMA INVOLVING INTRAPELVIC LYMPH NODES |


| D409 | Neoplasm of uncertain behavior of male genital organ, | |
|---|---|---|
| | unspecified | |
| D4100 | Neoplasm of uncertain behavior of unspecified kidney | |
| D4101 | Neoplasm of uncertain behavior of right kidney | |
| D4102 | Neoplasm of uncertain behavior of left kidney | |
| D4110 | Neoplasm of uncertain behavior of unspecified renal pelvis | |
| D4111 | Neoplasm of uncertain behavior of right renal pelvis | |
| D4112 | Neoplasm of uncertain behavior of left renal pelvis | |
| D4120 | Neoplasm of uncertain behavior of unspecified ureter | |
| D4121 | Neoplasm of uncertain behavior of right ureter | |
| D4122 | Neoplasm of uncertain behavior of left ureter | |
| D413 | Neoplasm of uncertain behavior of urethra | |
| D414 | Neoplasm of uncertain behavior of bladder | |
| D418 | Neoplasm of uncertain behavior of other specified urinary | |
| | organs | |
| D419 | Neoplasm of uncertain behavior of unspecified urinary organ | |
| - 1-2 | ,,,,, | |
| D420 | Neoplasm of uncertain behavior of cerebral meninges | |
| D421 | Neoplasm of uncertain behavior of spinal meninges | |
| D421<br>D429 | Neoplasm of uncertain behavior of meninges, unspecified | |
| D430 | Neoplasm of uncertain behavior of brain, supratentorial | |
| D430 | Neoplasm of uncertain behavior of brain, supratentorial | |
| D431<br>D432 | Neoplasm of uncertain behavior of brain, unspecified | |
| D432<br>D433 | Neoplasm of uncertain behavior of brain, unspecified Neoplasm of uncertain behavior of cranial nerves | |
| D434 | Neoplasm of uncertain behavior of spinal cord | |
| D438 | Neoplasm of uncertain behavior of other specified parts of | |
| | central nervous system | |
| D439 | Neoplasm of uncertain behavior of central nervous system, | |
| | unspecified | |
| D440 | Neoplasm of uncertain behavior of thyroid gland | |
| D4410 | Neoplasm of uncertain behavior of unspecified adrenal gland | |
| D4411 | Neoplasm of uncertain behavior of right adrenal gland | |
| D4412 | Neoplasm of uncertain behavior of left adrenal gland | |
| D442 | Neoplasm of uncertain behavior of parathyroid gland | |
| D443 | Neoplasm of uncertain behavior of pituitary gland | |
| D444 | Neoplasm of uncertain behavior of craniopharyngeal duct | |
| D445 | Neoplasm of uncertain behavior of pineal gland | |
| D446 | Neoplasm of uncertain behavior of carotid body | |
| D447 | Neoplasm of uncertain behavior of aortic body and other | |
| | paraganglia | |
| D449 | Neoplasm of uncertain behavior of unspecified endocrine | |
| | gland | |
| D45 | Polycythemia vera | |
| D460 | Refractory anemia without ring sideroblasts, so stated | |
| D461 | Refractory anemia with ring sideroblasts | |
| D4620 | Refractory anemia with excess of blasts, unspecified | |
| D4621 | Refractory anemia with excess of blasts 1 | |
| D4622 | Refractory anemia with excess of blasts 2 | |
| D464 | Refractory anemia, unspecified | |
| D469 | Myelodysplastic syndrome, unspecified | |
| D46A | Refractory cytopenia with multilineage dysplasia | |
| D46B | Refractory cytopenia with multilineage dysplasia and ring | |
| 55 | sideroblasts | |
| D46C | Myelodysplastic syndrome with isolated del(5q) | |
| D-10C | chromosomal abnormality | |
| D467 | · | |
| D46Z | Other myelodysplastic syndromes | |
| D470 | Histiocytic and mast cell tumors of uncertain behavior | |
| D471 | Chronic myeloproliferative disease | |
| D473 | Essential (hemorrhagic) thrombocythemia | |
| D479 | Neoplasm of uncertain behavior of lymphoid, hematopoietic | |
| | and related tissue, unspecified | 1 |


Drug abuse or dependence (includes alcohol)


Venous throm boem bolism


## Appendix A Comorbid conditions
